

| Protocol Number: | MC2-01-C6 | |
|---|---|---|
| Protocol Title: | A Multicentre, Open-label, Single-group Maximal Use Trial,<br>Evaluating the Safety and Pharmacokinetic Profile of the Active<br>Ingredients and their Metabolites after application of MC2-01 Cream<br>in Adolescent Subjects (age 12 to 16 years, 11 months) with Extensive<br>Psoriasis Vulgaris | |
| SAP version: | SAP for Interim Analysis Final 3.0 dated 07 September 2020 | |
| Effective date: | 07 September 2020 | |
| Reviewed and<br>Approved by | Johan Selmer | Chief Medical Officer, MC2 Therapeutics |
| | Date: | Signature: |
| Reviewed and<br>Approved by | Irene Sandholdt | Senior Project Manager, MC2 Therapeutics |
| | Date: | Signature: |
| Reviewed and<br>Approved by | Cathrin Baum | Project Manager, proinnovera GmbH |
| | Date: | Signature: |
| Reviewed and<br>Approved by | Leyla Tsakuginova | Lead Clinical Data Manager |
| | Date: | Signature: |
| Reviewed and<br>Approved by | Georgiy Smirnov | Head of Statistical Programming,<br>Data MATRIX |
| | Date: | Signature: |
| Prepared by | Kristina Bondareva | Head of Biostatistics Department,<br>Data MATRIX |
| | Date: | Signature: |



# **Revision History**

| No | Date | <b>Changes Implemented</b> | Version Number |
|---|---|---|---|
| 1 | 21JUL2020 | New document | 1.0 |
| 2 | 25AUG2020 | Updates for Finalization: List of laboratory parameters for analysis and corresponding units was corrected. Mistypes were corrected. | 2.0 |
| 2 | 07SED2020 | Updates after Data Review Meeting: Listing of Study Drug Accountability was added. Numbering of TFLs was updated. Minor changes in the TFLs shells were implemented. In Section 10 it was specified that Cmax is determined as maximum of the observed | 2.0 |
| 3 | 07SEP2020 | concentration values <b>after dosing</b> . | 3.0 |



## **Table of Contents**

| 1. Abbreviations and Definitions | |
|--------------------------------------------------|---|
| 2. Introduction | |
| 3. Study Objectives and Endpoints | |
| 3.1. Study Objectives | 6 |
| 3.2. Endpoints | 7 |
| 4. Study Design | 8 |
| 4.1. General Study Design and Plan | |
| 4.2. Randomization and Blinding | |
| 5. Sample Size | |
| 6. General Considerations. | |
| 6.1. Timing of Analyses. | |
| 6.2. Analysis Populations | |
| 6.3. Missing Data | |
| 6.4. Interim Analyses and Data Monitoring | |
| 6.5. Multi-center Studies | |
| 6.6. Multiple Testing | |
| 7. Summary of Study Data | |
| 7.1. Subject Disposition | |
| 7.2. Protocol Deviations | |
| 7.3. Demographic and Baseline Variables | |
| 7.4. Concurrent Illnesses and Medical Conditions | |
| 7.5. Prior and Concurrent Medications | |
| 7.6. Prior and Concurrent Procedures | |
| 8. Efficacy Analyses | |
| 9. Safety Analyses | |
| 9.1. Exposure | |
| 9.2. Adverse Events | |
| 9.3. Pregnancies | |
| 9.4. Clinical Laboratory Evaluations | |
| 9.5. Other Safety Measures | |
| 10. Pharmacokinetics | |
| 11. Other Analyses | |
| 12. Reporting Conventions | |
| 13. Technical Details | |
| 14. Summary of Changes to the Protocol | |
| 15. References | |
| 16. Listing of Tables, Listings and Figures | |
| 16.1. Tables | |
| 16.2 Figures | |
| 16.3. Listings | |
| Appendix 1. TFLs Shells | |
| Tables Shells | |
| Subject Disposition | |
| Protocol Deviations | |
| Demographic Characteristics | |
| Baseline Variables | |
| Medical HistoryPrior and Concomitant therapy | |
| ** | |
| Exposure | |
| Pharmacokinetics Analyses | |
| Adverse Events | |
| HPA Axis Suppression | |
| Calcium Metabolism | |
| Clinical Laboratory Evaluation | |
| Local Skin Reactions Assessment | |



| Vital signs | 83 |
|---------------------------------------------------|-----|
| Physical Examination | 88 |
| ECG | |
| Physician Global Assessment of Psoriasis Severity | |
| Body Surface Area Involvement Assessment | |
| Psoriasis Treatment Convenience Scale | 102 |
| Figures Shells | 104 |
| Listings Shells. | |

# 1. Abbreviations and Definitions

The abbreviations and the definitions used in this document are listed below.

| | d the definitions used in this document are listed below. |
|--------------|------------------------------------------------------------|
| Abbreviation | Definition |
| ACE | Angiotensin converting enzyme |
| ACTH | Adrenocorticotropic hormone |
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| AR | Adverse Reaction |
| AUC0-t | Area under the time-concentration curve from time |
| | zero to the last measurable concentration |
| AUC0-5 | Area under the time-concentration curve from time |
| | zero to 5 hours imputing the lower limit of quantification |
| | (LLoQ) for concentrations below LLoQ |
| BDP | Betamethasone dipropionate |
| BLQ | Below limit of quantification |
| BSA | Body surface area |
| CAL | Calcipotriene (United States term) / Calcipotriol |
| | (European Union term) |
| Cmax | Maximum plasma drug concentration |
| CRO | Contract Research Organisation |
| CSR | Clinical Study Report |
| CYP 3A4 | Cytochrome P450 3A4 |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| FDA | Food and Drug Administration |
| HPA | Hypothalamic-pituitary-adrenal |
| ICF | Informed consent form |
| ICH-GCP | International Conference on Harmonisation-Good |
| | Clinical Practice |
| IEC | Independent Ethics Committee |
| IP | Investigational product |
| IRB | Institutional Review Board |
| LLoQ | Lower Limit of Quantification |
| LSR | Local Skin Reactions |
| MCV | Mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MUsT | Maximal Usage Trial |
| OTC | Over the counter |
| PGA | Physician's Global Assessment |
| PK | Pharmacokinetics |
| PTCS | Psoriasis Treatment Convenience Scale |
| PTH | Parathyroid hormone |
| PUVA | Psoralen + ultraviolet A |
| RBC | Red blood cell |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SOP | Standard operating procedure |
| SUSAR | Suspected unexpected serious adverse reaction |
| SV1, SV2 | Screening Visit 1, Screening Visit 2 |
| Tmax | Time to maximum plasma drug concentration |



| US | United States |
|-----|------------------|
| UVB | Ultraviolet B |
| WBC | White blood cell |

#### 2. Introduction

This SAP is written according to ICH E9 Guideline [1] and Data MATRIX LLC SOP [2, 3] using the Protocol Final version 5.0 dated 23SEP2018 including Amendment dated 09JUN2020 and CRF Final version 1.2 dated 09JUL2020.

The purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis, described in the Protocol, and to include detailed procedures for executing the statistical analysis.

Based on FDA recommendation the trial is subject to a Temporary Halt, for non-safety reasons, to evaluate the study data in an interim analysis. It was decided to include data from all subjects who has been enrolled in the trial at the time of the interim analysis and perform analysis of all endpoints initially planned in the clinical study protocol.

This SAP needs to be finalized and signed prior to database lock for interim analysis and applies to the interim data analysis. Revisions to the approved SAP may be made prior to database lock for the interim analysis. In case of deviation from the finalized SAP, explanation will be provided in the clinical study report (CSR).

The interim report will be shared with FDA as post-approval supplement. Based on this report and subsequently feedback from FDA, it will be decided if the MC2-01-C6 study should be permanently closed or re-activated. In case the decision is made to resume the recruitment into the study, final statistical analysis will be conducted. A separate SAP will be prepared and finalized before the database lock for the final analysis.

#### 3. Study Objectives and Endpoints

## 3.1. Study Objectives

#### 3.1.1. Primary Objective

The primary objectives are to evaluate the effect of MC2-01 cream on the HPA axis and calcium metabolism following once daily topical application under maximum-use conditions in subjects with extensive psoriasis vulgaris.

#### 3.1.2. Secondary Objective

The secondary objective is to evaluate the pharmacokinetic profile of the active ingredients and their main metabolites following once daily topical application of MC2-01 cream under maximum-use conditions in adolescent subjects (age 12 to 16 years, 11 months) with extensive psoriasis vulgaris.



#### 3.2. Endpoints

#### 3.2.1. Primary Endpoint

#### HPA axis

Subjects with serum cortisol level of 18 µg/dL or less at 30 minutes after ACTH challenge test at Week 4 and Week 8.

#### • Calcium metabolism

Changes from Baseline to Week 4 and Week 8 in:

- Albumin-corrected serum calcium;
- Ratio of urinary calcium to creatinine\*.
- \*Spot analysis, second morning urine sample

## 3.2.2. Secondary Endpoints

• Plasma PK parameters (AUC0-t, AUC0-5, Cmax and Tmax) will be calculated at Week 4. The PK parameters AUC0-5 and Cmax will be calculated using standard formulas inserting the lower limit of quantification (LLOQ) for non-quantifiable levels of the analyte; therefore, AUC0-5 will be an upper limit in case at least one time-point shows a non-quantifiable level of the analyte, and Cmax will be an upper limit in case all time points show non quantifiable levels of the analyte. For a given analyte, the PK parameters AUC0-t and Tmax will be calculated if at least one time-point shows a quantifiable level of the analyte. The PK parameters will be summarised using appropriate descriptive statistics including median, lower and upper quartiles, minimum and maximum.

Blood samples for PK assessments will be collected at

- SV2 (baseline sample)
- Week 2 (single time point before application of IP)
- Week 4; before application of IP and then at 1, 3, and 5 hours after the application.
- Week 8; (single time point. Subject should not apply IP on the day of the Week 8 visit)

The samples will be assayed for concentrations of the active ingredients (BDP and CAL) and for their main metabolites; MC1080 and betamethasone 17-propionate, respectively.

#### 3.2.3. Safety Endpoints

- Adverse events (AEs) and serious adverse events (SAEs);
- Local skin reaction:
- Changes in safety laboratory test results;
- Changes in ECGs;
- Changes in vital signs and physical examinations.

#### 3.2.4. Other Endpoints

• The proportion of subjects with treatment success, defined as a minimum 2-point decrease from baseline in the PGA on the body (trunk and/or limbs), and with or without scalp at Week 4 and Week 8.



• Subject assessment of treatment convenience at Week 8 using a Psoriasis Treatment Convenience Scale.

## 4. Study Design

#### 4.1. General Study Design and Plan<sup>1</sup>

This is a phase 2, open-label, single-group, multicentre trial in which the investigational product (IP), MC2-01 cream, is investigated in adolescent subjects (age 12 to 16 years, 11 months) with clinically diagnosed extensive psoriasis vulgaris of at least moderate disease severity (according to the Physician's Global Assessment of Disease Severity; PGA) on body (trunk and/or limbs), and with or without scalp involvement.

After written informed assent is provided by the subject and written informed consent is provided by the parent(s) or legal guardian(s) and the consent document is signed by the investigator or designee the subjects will undergo screening procedures. For subjects requiring a washout period, informed assent/informed consent must be completed prior to washout. Prior to Screening Visit 2 (SV2) the subject (or the parent(s) or legal guardian(s)) is instructed to keep a diary for a 4-day registration of the daily intake of calcium-rich nutrients. At SV2, a second morning urine sample will be collected at the site for analysis of the urinary calcium excretion. Subjects will have their HPA axis function assessed and a baseline PK sample is collected along with other baseline assessments to confirm the subject's eligibility before Day 0/Visit 1.

Subjects who fulfil all inclusion and exclusion criteria at Day 0/Visit 1 are enrolled in the trial and will apply one dose of trial medication topically once daily for 8 weeks.

Please refer to Figure 1 for an overview of the trial design.

Trial subjects will be enrolled at approximately 12 sites in Europe.

At Week 4 and Week 8, the effect of once-daily use of MC2-01 cream on the HPA axis and the calcium metabolism will be evaluated. Other assessments (local skin reactions, AEs, laboratory tests, electrocardiogram (ECG), vital signs and physical examination) and efficacy assessments are also performed. At Week 4, the PK profile of calcipotriol (CAL), betamethasone dipropionate (BDP) and their main metabolites MC1080 and betamethasone 17-propionate, respectively, will be assessed.

#### Figure 1

<sup>&</sup>lt;sup>1</sup> This section is based on the sections 4.1 "Overall Trial Design.





<sup>\*</sup>There should be at least four days between SV1 and SV2 in order to keep the food diary for 4 days prior to SV2.

The maximum trial duration for each subject will be approximately 18 weeks and includes a screening period of up to 6 weeks (if washout of medication is required), a treatment period of 8 weeks, and a follow-up period of up to 4 weeks. After Week 8 (Visit 5) a follow-up visit is required for all subjects. The end of trial is defined as last subject last visit.

**Table 1** Schedule of Activities



| | SV 1 a | SV 2 | Visit<br>1 | Visit<br>2 | Visit 3 | Visit<br>4 | Visit<br>5 | Follow-<br>up<br>Visit <sup>b</sup> |
|---|---|---|---|---|---|---|---|---|
| | | | Day 0 | Week<br>2 | Week<br>4 | Week<br>6 | Week<br>8 | FU |
| Examination | Day - 42 to Day - 8 | Day<br>-7 to<br>- 4 | Day 0 | Day<br>14 ± 2 | Day 28 ± 2 | Day 42 ± 2 | Day 56 ± 2 | Day 70-<br>84 ± 2 |
| Informed assent/Informed consent c | X | | | | | | | |
| Inclusion/exclusion criteria | (X) | | X | | | | | |
| Urine pregnancy test <sup>d</sup> | X | | X | | | | | |
| Serum pregnancy test <sup>d</sup> | | X | | | X | | X | |
| Demographics, medical history | X | | | | | | | |
| Prior and concomitant medication | X | X | X | X | X | X | X | |
| Physical examination | X | | X | | X | | X | X |
| PGA | (X) | (X) | X | X | X | X | X | |
| Body Surface Area (BSA) involvement | (X) | (X) | X | | X | | X | |
| Vital signs | | | X | X | X | X | X | |
| Laboratory assessments | | X | | | X | (X)e | X | (X) |
| ACTH challenge test <sup>f</sup> | | X | | | X | | X | (X) |
| Morning urine assessment (second morning urine) | Instruct | X | | Instruct | Instruct<br>X | Instruct (X)g | Instruct<br>X | (X) |
| Review food diary | Instruct | X | | Instruct | Instruct<br>X | Instruct (X) <sup>g</sup> | Instruct<br>X | (X) |
| PK pre-dose blood sample (Single) | | X | Instruct | X | | Instruct | X | |
| PK serial blood samplesh | | | | Instruct | X | | | |
| 12-Lead ECG | | X | | | X | | X | |
| Psoriasis Treatment<br>Convenience Scale | | | | X | X | | X | |
| Dispense IP and diary for compliance | | | X | X | X | X | | |
| Collect IP | | | | X | X | X | X | |
| Compliance | | | | X | X | X | X | |
| Adverse event(s)i | | X | X | X | X | X | X | X |
| Local Skin Reactions | | | X | X | X | X | X | |

a) A washout period of up to 6 weeks must be completed if the subject has been treated with anti-psoriatic treatments or other relevant medication, as defined by exclusion criteria.

There should be at least four days between SV1 and SV2 in order to keep the food diary for 4 days prior to SV2. Items denoted in [brackets] must be reviewed during screening, to assess if the subject is otherwise eligible. Such items must be checked for any change in eligibility status at Visit 1/Day 0 after the washout is completed.

b) Follow-up visit is required 2 weeks after the Week 8 visit. For subject with HPA axis suppression at Week 8 the follow-up visit should be 4 weeks after the Week 8 visit.

If the albumin-corrected serum calcium or the urinary calcium creatinine ratio is elevated at Week 8 a repeat test should be performed. In case of a repeat of the urinary calcium creatinine ratio the subject should be instructed to record the calcium intact 4 days prior to the visit.

For Czech Republic and Hungary: if an on-site visit is not required the follow up visit can be a telephone call 2 weeks after Week 8 to ask for the wellbeing of the subject.

In addition, subjects discontinued due to a treatment-related AE will be monitored until the AE is resolved or until the medical condition of the subject is stable.

- c) Written informed assent must be provided by the subject and written informed consent must be provided by the parent(s), legal guardian(s) and the consent documents signed by the investigator or designee before any trial related procedures are carried out. For subjects requiring a washout period, informed assent/informed consent must be completed prior to washout.
- d) All female subjects.
- e) If serum albumin-corrected serum calcium is above the reference range at Week 4 a repeat test should be performed at Week 6.
- f) The ACTH challenge test must be performed between 7 and 9 AM, before IP application.
- g) If the urinary calcium: creatinine ratio is above the reference range at Week 4, a repeat test should be performed, and the food diary filled in at Week 6. If the repeat test is also above the reference range, 24-hour urine collection must be performed.
- h) Blood samples for PK analysis are drawn before IP application (pre-dose sample) and 1, 3, and 5 hours after IP application.
- i) AEs are to be collected from the date of signing informed assent/informed consent and first trial-related activity is performed.

## 4.2. Randomization and Blinding<sup>2</sup>

This is an open-label trial. All subjects who fulfil the trial eligibility requirements will be assigned to treatment with MC2-01. Neither randomization nor blinding will be performed.

<sup>&</sup>lt;sup>2</sup> This section is based on the section 6.5 "Assignment to Treatment" of clinical study Protocol.



## 5. Sample Size<sup>3</sup>

It is planned to enroll approximately 30 subjects. The choice of sample size in this trial is based on regulatory considerations with respect to common practice in maximum use studies. For the PK population, the aim is to have at least 20 subjects included that have at least completed Week 4 (Visit 3).

The choice of sample size in this trial is not based on statistical considerations, but rather on regulatory considerations with respect to common practice in maximum use studies evaluating pharmacokinetic profiles and evidence of HPA safety.

#### 6. General Considerations

#### 6.1. Timing of Analyses

One interim analysis following study completion by 7 treated subjects will be prepared.

The final analysis will be prepared in case the MC2-01-C6 is re-activated (refer to Section 6.4).

#### 6.2. Analysis Populations

The main subject samples of interest are defined as follows.

The 'All enrolled subjects': all subjects for whom Informed Consent/Assent were obtained:

The 'Allocated to treatment': all subjects for whom Informed Consent/Assent were obtained and who had successfully completed Screening procedures and to whom any amount of trial medication was dispensed.

The 'Safety population': all subjects who are enrolled in the trial and dispensed the trial medication at Visit 1/Day 0, excluding subjects who return all of the trial medication unused. The Safety population will be used for all safety analyses other than evaluation of the HPA-axis.

The 'PK population': all subjects in the Safety population who have received the planned application of treatment at the Week 4 visit and have had at least one blood draw for PK assessment at Week 4.

The 'HPA population': all subjects in the Safety population that show normal HPA function at SV2:

• Serum cortisol concentration above 4.5mcg/dl (160nmol/l) before ACTH-challenge and equal or above 18 mcg/dl (500 nmol/l) 30 minutes after ACTH challenge, at SV2.

The HPA population will be used for the HPA axis suppression analysis.

CONFIDENTIAL AND PROPRIETARY Data MATRIX Ltd.

<sup>&</sup>lt;sup>3</sup> This section is based on the section 5.1 "Subject Population" and 8.2 "Sample Size and Power Considerations" of clinical study Protocol.



For interim analyses *Interim* < Population Name > will be used for reporting.

#### 6.3. Missing Data

No imputation will be made for missing data apart from missing or partial adverse event start date and concomitant medication end date necessary to calculate the treatment-emergent and prior/concomitant/post-treatment flags, correspondingly.

If the information about end date for prior/concomitant therapy is missing or incomplete, the following rules (Table 2.1.1 and Table 2.1.2) will be used for the classification of therapy as prior, concomitant or post-treatment.

Table 2.1.1 Management of partial and missing prior/concomitant therapy start date.

| Day | Month | Year | Processing |
|---|---|---|---|
| | | | Therapy will be classified as post- |
| | | | treatment, if start month and year > |
| is missing | is known | is known | month and year of the last IMP dose, |
| | | | else – as prior or concomitant according |
| | | | to the definition and Table 2.1.2 |
| is missing | is missing | is known | Therapy will be classified as post- |
| | | | treatment, if start year > year of the last |
| :- 1 | is missing | is known | IMP dose, else – as prior or |
| is known | | | concomitant according to the definition |
| | | | and Table 2.1.2 |
| is missing | is known | is missing | Therapy will be classified as prior or |
| is known | is missing | is missing | concomitant according to the definition |
| is missing | is missing | is missing | and Table 2.1.2 |

Table 2.1.2 Management of partial and missing prior/concomitant therapy end date.

| Day | Month | Year | Processing |
|---|---|---|---|
| is missing | is known | is known | Therapy will be classified as prior, if end month and year < month and year of the first IMP dose, else – as concomitant |
| is missing | is missing | is known | Therapy will be classified as prior, if |
| is known | is missing | is known | end year < year of the first IMP dose,<br>else – as concomitant |
| is missing | is known | is missing | Thereny will be elegated as |
| is known | is missing | is missing | Therapy will be classified as concomitant |
| is missing | is missing | is missing | Conconntant |

The medical history records will be categorized in prior/concurrent categories in a similar way.



If the information about adverse event start date and time is missing or incomplete, the following rules (Table 2.2) will be used for the classification of adverse events as TEAEs and non-TEAEs (occurred before the start of study treatment) and for identification of TEAEs occurred up to Week 4.

Table 2.2 Management of partial and missing AE start date.

| Day | Month | Year | TEAE flag | Occurrence up to Week 4 |
|---|---|---|---|---|
| is<br>missing | is<br>known | is<br>known | AE will be classified as TEAE, if month and year ≥ month and year of the first dose of study therapy | TEAE will be classified as occurring up to Week 4, if month and year <= month and year of the Visit 3 / Week 4 or subject discontinued before Visit 3 / Week 4 |
| is<br>missing | is<br>missing | is<br>known | AE will be classified as | TEAE will be classified as occurring up to Week 4, if year <= year of the |
| is known | is<br>missing | is<br>known | TEAE, if year ≥ year of the first dose of study therapy | Visit 3 / Week 4 or subject discontinued before Visit 3 / Week 4 |
| is | is | is | | TEAE will be classified as occurring |
| missing | known | missing | | up to Week 4 |
| is known | is | is | AE will be classified as | |
| 15 KHOWH | missing | missing | TEAE | |
| is | is | is | | |
| missing | missing | missing | | |

Original dates (without imputation) will be used for data listings.

## 6.4. Interim Analyses and Data Monitoring<sup>4</sup>

Based on FDA recommendation the trial will be subject to a Temporary Halt to evaluate the study data in an interim analysis and create an interim report.

The interim report will be shared with FDA as post-approval supplement. Based on this report and subsequently feedback from FDA, it will be decided if the MC2-01-C6 study should be permanently closed or re-activated.

Interim analysis will be conducted on complete data from all subjects who had been enrolled into the trial at the time of interim analysis. Interim analysis will include the analysis of all endpoints initially planned in the clinical study protocol.

#### 6.5. Multi-center Studies

Data from all centers will be merged and analyzed as one population for all study endpoints.

#### 6.6. Multiple Testing

No adjustment for multiplicity is planned.

<sup>&</sup>lt;sup>4</sup> This section is based on the section 8.11 "Interim analysis" of clinical study Protocol including Amendment.



### 7. Summary of Study Data

Demographic and other baseline characteristics and safety data will be summarized by time point of assessment and listed.

## **Default Summary Statistics**

The default summary statistics for quantitative and ordinal variables will be the number of observations (n), mean, standard deviation (SD), median, minimum (Min) and maximum (Max).

### **Default Frequency Tabulations**

For qualitative variables, the number and percentage (n, %) of subjects with non-missing data per category and total number of subjects with non-missing data where applicable will be the default summary presentation.

For AEs, medical history, concomitant medications and protocol deviations, however, the denominator for the percentage calculation will be the number of subjects in the corresponding population.

The number of decimals for each descriptive statistic will be determined by the following rules:

- mean, median: +1 decimal symbols compared to the analyzed variable values;
- standard deviation: +1 decimal symbols compared to the analyzed variable values;
- first (Q1) and third (Q3) quartiles: +1 decimal symbols compared to the analyzed variable values;
- minimum and maximum values: the same as for the analyzed variable values;
- percentages will be rounded to one decimal symbol;
- confidence intervals will be presented with accuracy of the estimated value.

The maximum number of decimal places in the statistical report is four. If some descriptive statistic has more than four decimal places after above mentioned rules application, this value will be rounded to four decimal places.

#### Statistical Tests and Common Calculations

Unless otherwise specified in the description of the analyses, the following arrangements will be applied:

- 95% two-sided confidence intervals (CI);
- CIs for mean values will be calculated based on normal distribution (SAS procedure UNIVARIATE with CIBASIC option);
- CIs for proportions will be computed using the exact (Clopper-Pearson) method.

For descriptive statistics, the following rules will be applied:

- "<X.XX" results (e.g. below the limit of quantification, BLQ) for safety laboratory parameter values will be imputed with numeric result calculated as X.XX – 0.01. The number to be subtracted will be defined based on number of decimal places in observed values (e.g., if number of decimal places is 0 subtract 1, if number of decimal places is 1 subtract 0.1, etc.). Imputed data will be used in summaries and calculations, but original</p>



result will be listed.

For quantitative measurements, changes from baseline will be calculated as [value at post-baseline visit X – baseline value].

The baseline value for a variable in common cases is defined as the last non-missing value collected before the first study drug application.

Study day for each event will be calculated from the reference start date (date when subject was first exposed to study drug).

If the date of the event is on or after the reference date, then

$$study day = (date \ of \ event - reference \ date) + 1.$$

If the date of the event is prior to the reference date, then

$$study day = (date \ of \ event - reference \ date).$$

For partial dates study day will not be calculated.

The following visit windows were defined in the clinical study protocol:

| Visit Name | Visit Short<br>Name | Anchor | Target<br>Day | First day of<br>the visit<br>window | Last day of<br>the visit<br>window |
|---|---|---|---|---|---|
| Screening Visit 1 | SV1 | First application | - | -42 | -8 |
| Screening Visit 2 | SV2 | First application | - | -7 | -4 |
| Visit 1 (Day 0) | V1 (Day 0) | First application | 1 | 1 | 1 |
| Visit 2 / Week 2 | V2/Week 2 | First application | 15 | 13 | 17 |
| Visit 3 / Week 4 | V3/Week 4 | First application | 29 | 27 | 31 |
| Visit 4 / Week 6 | V4/Week 6 | First application | 43 | 41 | 45 |
| Visit 5 / Week 8 | V5/Week 8 | First application | 57 | 55 | 59 |
| Follow-up Visit | FU | Last application | 15 | 13 | 17 |

Assessments performed out of the planned visit windows will be assigned to the nearest of the surrounding planned visits if there is no valid result from a planned assessment for this visit. If assessments at both surrounding visits are missing and they are equidistant, the assignment is performed to the later one. Otherwise the assessments will not be included in summaries and will be listed only.

Unscheduled and early termination visit assessment can be assigned to the planned visit in a similar manner. Unscheduled assessment can also be used in the derivations such as baseline or most extreme post-baseline assessments. All assessments including unscheduled should be presented by subject in the data listings.

### 7.1. Subject Disposition

The following disposition summaries will be provided:

- A summary of the number of subjects who provided the informed consent / informed assent, the number of screen failures (including those subjects who satisfied the inclusion/exclusion criteria but for whom no study drug was dispensed) with reasons for premature study termination
- A summary of the number of screen failure subjects violated any inclusion/exclusion criterion,



by criterion

- A summary of the number of subjects allocated to treatment, the number and percentage of subjects attended each study visit (Allocated to treatment set)
- A summary of the number and percentage of subjects included in each population for statistical analysis (Allocated to treatment set)
- A summary of the number and percentage of subjects completed the study and prematurely discontinued from the study by reason for study discontinuation (Allocated to treatment set)
- A summary of the number and percentage of subjects completed the study treatment and prematurely discontinued the study treatment before Week 8 visit by reason for discontinuation (Safety population).

By-patient listings of disposition details will be provided for all enrolled subjects.

#### 7.2. Protocol Deviations

Number and percentage of subjects with at least one protocol deviation and at least one major protocol deviation will be tabulated by category and subcategory and overall (Allocated to treatment set). All protocol deviations will be listed (All Enrolled subjects).

Major protocol violations include but are not limited to:

- Informed consent not received or provided after the first study visit;
- Inclusion/exclusion criteria violations in subjects allocated to treatment;
- Use of prohibited concomitant medication or non-drug therapy that may affect study results or their interpretation;
  - Week 4 assessments performed more than 14 days after the scheduled date;
  - Week 8 assessments performed more than 14 days after the scheduled date;

Major protocol violations will be finalized and approved by MC2 at the data review meeting.

## 7.3. Demographic and Baseline Variables

eCRF form: "DEMOGRAPHICS", "VITAL SIGNS".

Descriptive statistics for the following demographic, anthropometric and other baseline characteristics will be presented in accordance with section 7:

- demographic characteristics: country, age, gender, race, ethnic origin;
- anthropometric characteristics: height (cm), weight (kg), body mass index (BMI, kg/m<sup>2</sup>);



eCRF form: "FITZPATRICK SKIN TYPE ASSESSMENT", "BODY SURFACE AREA INVOLVEMENT ASSESSMENT", "PHYSICIAN'S GLOBAL ASSESSMENT OF PSORIASIS SEVERITY", "MAIN DIAGNOSIS", "LOCAL SKIN REACTIONS ASSESSMENT".

- Fitzpatrick skin type;
- Scalp BSA psoriatic involvement (%), Neck, Trunk and/or Limbs BSA psoriatic involvement (%), Total psoriatic involvement (%);
- Physician's Global Assessment of psoriasis severity (PGA);
- Duration of disease (months);

Specific calculations and/or conversions include but are not limited to the following:

Body mass index will be calculated as weight  $(kg) / [height (m)]^2$ .

Duration of disease will be calculated in months as (date of informed consent - date of diagnosis + 1) / 30.4375. In order to calculate disease duration partial diagnosis date will be imputed with 15th day of the same month, if month and year of diagnosis are collected. If only year of diagnosis is collected, diagnosis date will be imputed as July 1<sup>st</sup> of the corresponding year. If the imputed date of diagnosis is later than the date of informed consent, the date of informed consent will be used.

All data will be listed.

#### 7.4. Concurrent Illnesses and Medical Conditions<sup>5</sup>

eCRF form: "MEDICAL HISTORY"

Medical history findings will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 22.0 (or more recent version if available) according to Data MATRIX SOP [4], and will be presented by Primary System Organ Class (SOC) and Preferred Term (PT) within SOC.

Prior and concurrent diagnoses will be tabulated separately.

Medical history findings will be reported on a by-patient basis. This implies that if the subject suffered the same event (mapped to same PT) repeatedly the event will be counted once and only once for appropriate PT. Within SOC subjects may have reported more than one PT. The SOCs and PTs within each SOC will be sorted in descending order of total incidence.

Classification of condition/diagnosis as either Prior or Concurrent will be based on stop date of condition/diagnosis in "MEDICAL HISTORY" eCRF form. The number (%) of subjects reporting any medical history will be presented in tables by SOC and PT.

Medical history records with stop date prior to the date of first dose of study therapy will be classified as Prior conditions/diagnoses. If a condition/diagnosis stops on or after the date of first

\_

<sup>&</sup>lt;sup>5</sup> This section is based on the section 7.1 "Demographics and Medical History" of clinical study Protocol.



dose of study therapy or is ongoing at the end of clinical study, then the condition/diagnosis will be classified as Concurrent. If the information about stop date of condition/diagnosis is missing or incomplete, the rules from section 6.3 will be applied for classification. Medical history record will be assumed to be Concurrent, unless there is clear evidence (through comparison of partial dates) to suggest that the condition/diagnosis stopped prior to the first dose of study therapy. If there is clear evidence to suggest that the condition/diagnosis stopped prior to the first dose of study therapy, the condition/diagnosis will be assumed to be Prior.

All data will be listed.

#### 7.5. Prior and Concurrent Medications<sup>6</sup>

eCRF form: "PRIOR/ CONCOMITANT THERAPY AND NON-DRUG THERAPY".

All medications, including OTC drugs, herbals, vitamins, dietary supplements etc., taken within 30 days prior to the start of the trial will be recorded at Screening (SV1 and/or SV2). Thereafter, a record of all medications and supportive therapy taken during the trial will be made.

All prior and concomitant medications (including non-drug therapy) will coded using the World Health Organization Drug Dictionary (WHODD) version B2 September 2018 (or more recent version if available) according to Data MATRIX SOP [4]. The number (%) of subjects reporting the use of any prior or concomitant medication will be presented in tables by pharmacological subgroup (3rd level) and chemical substance (5th level). Post-treatment medications will be reported in listing only.

Classification of treatment as either Prior, Concomitant or Post-Treatment will be based on start and stop date of medication in "PRIOR/CONCOMITANT THERAPY AND NON-DRUG THERAPY" eCRF form.

Medications that stop prior to the date of first dose of study therapy will be classified as Prior medications. If a medication stops on or after the date of first dose of study therapy (or "ONGOING") then the medication will be classified as Concomitant unless the medication started after the date of last IMP administration in which case it will be classified as Post-Treatment. If the information about stop date of medication is missing or incomplete, the rules from section 6.3 will be applied for classification. Medications will be assumed to be concomitant, unless there is clear evidence (through comparison of partial dates) to suggest that the medication stopped prior to the first dose of study therapy or started after the last dose of study therapy. If there is clear evidence to suggest that the medication stopped prior to the first dose of study therapy, the medication will be assumed to be Prior. If there is clear evidence to suggest that the medication started after the last dose of study therapy, the medication will be assumed to be Post-Treatment. By-patient listings will be provided with appropriate flagging of prior, concomitant and post-treatment records.

<sup>&</sup>lt;sup>6</sup> This section is based on the section 7.2 "Prior and Concomitant Medication" of clinical study Protocol.



#### 7.6. Prior and Concurrent Procedures

eCRF form: "PRIOR/ CONCOMITANT PROCEDURES".

Procedures will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 22.0 (or more recent version if available) according to Data MATRIX SOP [4].

All procedures recorded will be listed.

#### 8. Efficacy Analyses

Not Applicable.

#### 9. Safety Analyses

## **9.1.** *Exposure*<sup>7</sup>

Exposure and compliance will be evaluated based on the information from the "STUDY DRUG APPLICATION", "STUDY DRUG COMPLIANCE", "STUDY DRUG ACCOUNTABILITY", "END OF TREATMENT", "MISSING DOSES" eCRF form.

Subjects are to apply the IP topically once daily, preferably in the evening, for 8 weeks. The subject should apply enough IP to treat the entire affected areas and rub in gently to ensure that the plaques are saturated with the medication. Up to 3 tubes of 60 gram will be dispensed for a treatment period of two weeks including the allowed visit window of 2 days.

Only affected areas are to be treated. The subjects should therefore not continue treatment on a skin area which has been cleared but treatment may be restarted in case of recurrence at the subjects' discretion.

Dose modification can only occur after Week 4.

Subjects classified as clear at any of the on-treatment visits may stop the IP treatment at the investigator's discretion. They should remain in the trial and attend all visits up to and including the follow-up visit. The IP will continue to be dispensed to the subject, and IP treatment may be restarted at the subject's discretion. The subject should not discontinue treatment themselves between visits but is only allowed to stop using the IP treatment on the advice of the investigator at a scheduled visit.

The total duration of exposure is defined as the time interval in days between the first dose and the last dose, inclusive, of study drug as [(date of last dose – date of first dose+1)].

Total dose (g) administered during the study will be assessed based on study drug accountability data as [average weight of tube dispensed –weight of tube returned] summed over all tubes dispensed except for tubes assessed as unused or used but lost which will not be taken into account in the calculation. Average dispense weight is 75.54 g.

<sup>&</sup>lt;sup>7</sup> This section is based on the section 6.2 "Dosing Regimen" and 6.3 "Dose Modification" of clinical study Protocol.



Average weekly dose (g) will be calculated as [total dose (g) / (total duration of exposure / 7)].

Compliance will be estimated as [100% \* (number of required days in the time period assessed – number of missed doses during the time period assessed)/ number of required days in the time period assessed]. The number of required days is the total number of days between the first and the last application in the time period assessed excluding days with approved IMP discontinuation.

If a dose is missed due to approved discontinuation at a given day this day will not be included in the calculation of compliance. The period of time between the approved discontinuation at a scheduled visit and treatment restart (not inclusive) will not be taken into account in the calculation of compliance.

Treatment compliance will be categorized to less than 80% versus 80% or more.

Extent of exposure (days) will be calculated as [number of required doses - total number of missed doses]. The number of required doses is the total number of days between the first and the last application in the time period assessed excluding days with approved IMP discontinuation.

Number of missed doses will be summarized for subjects with at least one missed dose as a continuous variable, both using zero counts for those subjects from Safety Population who have not reported any missed dose and providing summary only for those subjects who reported at least one missed dose.

Total duration of exposure (days), total dose (g), weekly dose (g), treatment compliance (%), extent of exposure (days), number of missed doses will be summarized by time period (up to Week 2, up to Week 4 and Week 4 to Week 8) and for the entire treatment period to the Week 8 visit, using descriptive statistics in the Safety population.

The periods that the kits were used as recorded on "STUDY DRUG ACCOUNTABILITY" eCRF form will be used to assign the kit to one of the time periods for calculation of total dose (g) administered during each period (up to Week 2, up to Week 4 or Week 4 – Week 8). If the use period starts at Week 4 or Week 6 visit the time period is Week 4 to Week 8, if the use period starts before Week 2 (Week 4) and ends on or before Week 2 (Week 4), the time period is up to Week 2 (Week 4), otherwise time period cannot be determined.

The periods' start and end date will be defined through the actual dates of subject's visits. Week 2 (Week 4) visit date will be considered the last day of Week 0 – Week 2 (Week 4) period.

All exposure data will be listed by study period.

#### 9.2. Adverse Events

eCRF form: "ADVERSE EVENTS".

All registered AEs will be coded using the MedDRA version 22.0 (or a later version if available).

Treatment-emergent AEs will be summarized by the overall incidence of at least one event, incidence by body system, and incidence by body system and preferred term. Each subject will contribute only once (e.g., the first occurrence) to each of the rates, regardless of the number of occurrences (events) the subject experiences. Treatment-emergent AEs will be summarized by



severity (mild, moderate, or severe), and by relationship to trial product (none, possible, probable, or definite). An AE is treatment-emergent if its date of onset is on or after the date of the first application of the IP.

Only treatment emergent AEs will be summarized. In the listings, however, all occurrences of the AEs will be presented.

Number (percentage) of subjects and number of AEs will be presented for the Safety population in the following tables:

- All treatment-emergent AE / SAE;
- Treatment-emergent AE / SAE related to the study drug (relationship to trial product assessed by the investigator as possible, probable, or definite including those events where assessment is missing);
- TEAE by maximum severity;
- TEAE by closest relationship to study drug;
- TEAE related to study drug by maximum severity;
- TEAE related to cosyntropin;
- TEAE related to study procedures;
- TEAE leading to the permanent discontinuation of study drug (Action taken with IP="Drug withdrawn");
- TEAE leading to withdrawal (Did subject withdraw due to this AE?="Yes");
- TEAE leading to death (Outcome = "Death");
- Non-serious TEAEs that occurred at a frequency of >= 5% (if no events occurred at the 5% threshold all non-serious TEAEs will be tabulated).

This set of tables will be repeated for the adverse events occurring up to Visit 3 / Week 4. Treatment-emergent adverse events with start dates on or prior to Visit 3 / Week 4 date will be summarized separately. If subject discontinued from the study prior to Visit 3 / Week 4 his/her adverse events will also be included in these summaries. If subject missed Visit 3 / Week 4 the planned date of visit (study day) will be used to subset the events occurring up to Week 4.

Tables of TEAEs by maximum severity (closest relationship to study drug) will be prepared using the following rules: each SOC / PT category will include only the AEs with the worst severity (closest relationship) for each subject. In the Overall category, all AEs of the subjects will be presented. Each subject will be counted only once with the worst severity (closest relationship) in each SOC and each PT level as well as in the Overall level.

In case if severity or relationship to study drug is missing, the worst case value will be assumed and used in the summary.

All AEs/SAEs will be listed. Non-treatment emergent adverse events will be identified accordingly in the listing. Discontinuations from the trial due to AEs and SAEs will be listed by subject.



#### 9.3. Pregnancies

eCRF form: "URINE PREGNANCY TEST", "SERUM PREGNANCY TEST".

All female subjects will undergo a routine urine pregnancy test at SV1 and V1 (Day 0) and a serum pregnancy test at SV2, Week 4 & Week 8 as specified in the visit schedule (Table 1).

The results of these tests and pregnancies episodes will be reported in the listing.

#### 9.4. Clinical Laboratory Evaluations

eCRF form: "LABORATORY ASSESSMENT", "SERUM CHEMISTRY", "MORNING URINE ASSESSMENT", Central laboratory data.

Clinical laboratory data will be summarized by presenting shift tables using extended normal ranges (baseline to most extreme post-baseline value), by presenting summary statistics of raw data and change from baseline values (means, medians, standard deviations (SDs), ranges), and by the flagging of notable values (out of range values) in data listings.

Clinical laboratory evaluations as scheduled in the Table 1 include the following parameters:

- Hematology: hemoglobin, hematocrit, red blood cell (RBC) count, mean corpuscular volume (MCV), white blood cell (WBC) count, including differential count and platelet count.
- Serum biochemistry: cortisol, urea, glucose, creatinine, calcium, albumin, calcium (albumin corrected), sodium, potassium, chloride, phosphate, alkaline phosphatase (ALP), plasma parathyroid hormone (PTH).
  - 25-OH Vitamin D, only at SV2
- Morning urine assessment: calcium, phosphate, creatinine, volume, total calcium excretion, total phosphate excretion, total creatinine excretion, urinary calcium:creatinine ratio, urinary phosphate:creatinine ratio.
- Week 4: If albumin-corrected serum calcium is above the reference range at Week 4, a repeat test should be performed at Week 6. If the morning urinary calcium:creatinine ratio is above the reference range at Week 4, a repeat test should be performed at Week 6.
- Week 8: If the albumin-corrected serum calcium is above the reference range at Week 8, a repeat test is required 14 days ( $\pm$  2 days) after at a follow-up visit. If the urinary calcium:creatinine ratio is above the reference range at Week 8, a repeat test is required at a follow-up visit 14 days ( $\pm$  2 days) after Week 8. If the calcium-creatinine ratio is above the reference range at two consecutive visits during the trial, 24-hour urine collection must be performed.

For laboratory parameters the following tables will be presented according to section 7:

 descriptive statistics of measured values and changes from baseline by visit including highest/lowest post-baseline value;



- shift tables based on comparison with normal range (Low/Normal/High) by visit and to highest/lowest post-baseline value;
- frequency tables for Out of range: Normal/Out of range (Low/High) for laboratory parameters by visit.

Clinical laboratory values will be reported as complete listings of individual subject data.

A separate listing will be prepared for all clinically significant abnormal results.

## 9.5. Other Safety Measures

#### **HPA-axis suppression**

The primary outcome variable for HPA axis is serum cortisol level of less than 18  $\mu$ g/dL (500 nmol/L) at 30 minutes after ACTH challenge test (at Week 4 and Week 8).

The number and proportion of subjects with HPA-axis suppression at Week 4 and Week 8 will be summarised using frequency counts, percentages and exact 95% CI. Percentage will be calculated based on number of valid measurements (number of subjects for whom ACTH challenge test was performed) at each post-baseline visit. Number and proportion (95% CI) of subjects for whom HPA-axis suppression was noted at least once during the study will be presented. For Week 8, number and proportion of subjects with HPA-axis suppression will be additionally presented by HPA suppression status at Week 4.

Serum cortisol level at each time point (pre- and post- ACTH challenge test) will be summarized in tables with standard descriptive statistics for continuous variables and 95% CI for the means.

#### Calcium metabolism

Changes from Baseline to Week 4 and Week 8 in:

- Albumin-corrected serum calcium;
- Ratio of urinary calcium to creatinine\*.

\*Spot analysis, second morning urine sample

Descriptive statistics for measured parameters as well as changes from baseline will be presented by visit of assessment as scheduled in the Table 1.

#### Vital signs

eCRF form: "VITAL SIGNS".



Blood pressure and pulse rate will be taken with the subject in the sitting position with approximately 5 minutes' rest prior to measurement. Body temperature (oral or ear) will be also be measured.

Vital signs (pulse rate (beats/minute), and systolic and diastolic blood pressure (mm Hg), and oral or tympanic temperature (°C)), body weight (kg), body height (cm) and BMI (kg/m2) results will be presented in accordance with section 7.

Vital signs results will be presented by visit of assessment as scheduled in the Table 1.

Notable ranges are defined for vital signs according to Table 3.1. Notable values are post-baseline values outside the notable ranges, whether above or below, and are indicated as *notably abnormal*.

Table 3.1: Definition of Notable Ranges of Vital Signs

| Parameter | Notable Values and Changes from Baseline |
|---|---|
| Systolic blood | 90 mmHg or lower and decreased by 20 mmHg or more, |
| pressure | 180 mmHg or greater and increased by 20 mmHg or more |
| Diastolic blood | 50 mmHg or lower and decreased by 15 mmHg or more, |
| pressure | 110 mmHg or greater and increased by 15 mmHg or more |
| Pulse rate | 50 bpm or lower and decreased by 15 bpm or more, 120 bpm or greater and increased by 15 bpm or more |
| | 120 opin of greater and increased by 13 opin of more |

Normal ranges are defined for vital signs according to Table 3.2.



Table 3.2: Definition of Normal Ranges of Vital Signs

| Parameter | Units of | Age | | | Normal Ranges | |
|---|---|---|---|---|---|---|
| | Measure | Any | Low High | | | |
| | | | | | Low | High |
| Systolic blood pressure | mmHg | - | 12 | 17 | 80 | 160 |
| Diastolic blood pressure | mmHg | - | 12 | 17 | 50 | 100 |
| Pulse rate | Beats/min | - | 12 | 17 | 50 | 100 |
| Oral temperature | °C | _ | 12 | 17 | 35.0 | 37.5 |
| Tympanic temperature | °C | - | 12 | 17 | 35.0 | 37.5 |

Vital signs and body weight results will be presented as the following outputs:

- descriptive statistics for measured values and changes from baseline (vital signs, body weight, body height, BMI) by visit and highest/lowest post-baseline assessment (vital signs);
- frequency table for Out of range values, including frequency of Low and High values by visit and at any post-baseline assessment (vital signs);
- frequency table for notably abnormal values and changes from baseline (systolic blood pressure, diastolic blood pressure, pulse rate) by visit and at any post-baseline assessment.

All data will be listed. Notable values will be flagged.

#### **ECG**

#### eCRF form "ELECTROCARDIOGRAM".

A 12-lead ECG will be recorded at visits indicated in Table 1. Recording will take place after 5 minutes' rest in supine position. Recordings will be promptly transmitted to the central ECG vendor for interpretation. Additional (unscheduled) ECGs can be recorded for safety reasons at any time based on the judgement of the investigator.

Heart rate (beats/min), RR interval (msec), PR interval (msec), QRS duration (msec), QT interval (msec), QTC-B interval (msec) will be summarized using standard descriptive statistics for continuous variables in accordance with section 7.

Notable ranges are defined for electrocardiogram according to Table 4. Notable values are post-baseline values outside the notable ranges and are indicated as *notably abnormal*.



Table 4: Definition of Notable Ranges of ECG

| Parameter | Notable Values and Changes from Baseline |
|-----------|-----------------------------------------------|
| QTc | QTc interval > 450 msec |
| | QTc interval > 480 msec |
| | QTc interval > 500 msec |
| | QTc interval increases from baseline >30 msec |
| | QTc interval increases from baseline >60 msec |

A 12-lead electrocardiogram (ECG) results will be presented in accordance with section 7 by visit of assessment as scheduled in the Table 1 as the following outputs:

- frequency table for Normal/Abnormal clinically significant (Abnormal CS) / Abnormal non-clinically significant (Abnormal NCS) evaluation for General assessment (Total assessment) by visit and any post-baseline Abnormal and clinically significant Abnormal assessment;
- frequency table for notably abnormal values and changes from baseline (QTC-F interval, msec; QTC-B interval, msec) by visit and any post-baseline notably abnormal value;
- descriptive statistics of ECG parameters and their changes from baseline (Heart rate, beats/min; RR interval, msec; PR interval, msec; QRS duration, msec; QT interval, msec; QTC-F interval, msec; QTC-B interval, msec) by visit and highest/lowest post-baseline value.

All ECG data will be listed. Notable values will be flagged.

#### Physical examinations

eCRF form: "PHYSICAL EXAMINATION".

An abbreviated physical examination including general appearance, regional lymph nodes and a complete dermatological examination of the skin must be performed as scheduled in the Table 1.

Physical examination / dermatological examination results will be presented in accordance with section 7 by visit of assessment as the following output:

frequency table for Normal/Abnormal clinically significant (Abnormal CS) / Abnormal non-clinically significant (Abnormal NCS) evaluation.

All physical examination / dermatological examination data will be listed.



#### Local skin reactions

The local skin reaction assessment involves signs assessed by the investigator or designee and symptoms reported by the subject.

The investigator will assess the treatment area and/or immediate surrounding for the following identified signs:

- Perilesional erythema, scaling, edema, atrophy, vesicles and erosion/ulceration;
- Lesional vesicles, and erosion/ulceration.

The intensity of each local skin reaction category is to be graded according to the scale provided in Table 7-4 of the protocol. The most severe intensity observed for each category of the local skin reaction assessment is to be recorded.

Local skin reactions (LSR) sum score is defined as the sum of intensity grades across all areas and signs per visit. Per sign, the most intense reaction is defined as the maximum intensity grade across visits.

The subject will assess burning and pain after application. The investigator or designee will explain the scores provided in Table 7-4 of the Protocol and the subject will tell which one to mark.

The local skin reaction assessment results will be presented in accordance with section 7 as the following outputs:

- frequency table for investigator assessment of lesional/perilesional area and subject's assessment of burning and pain after application by visit of assessment as scheduled in the Table 1 and most severe post-baseline assessment;
- shift table from baseline to each post-baseline visit value and most severe post-baseline value;
- descriptive statistics of LSR sum scores and their changes from baseline for lesional/perilesional area by visit

#### 10. Pharmacokinetics

Samples for PK analysis will be collected through an untreated area of the skin, at the following time points:

- SV2: single time point
- Week 2 visit: single time point before IP application
- Week 4 visit: before the planned IP application at the visit and then at 1, 3, and 5 hours after the application
- Week 8 visit: single time point. Subject should not apply IP on the day of the Week 8 visit Subjects are to be instructed to apply their daily dose of IP in the morning on the day before the Week 2, Week 4 and Week 8 visits. On the day of these visits, the subjects should not apply any



IP before the visit. A reminder to the subject may be needed a few days before the scheduled visit.

The samples will be assayed for concentrations of the active ingredients (BDP and CAL) and for their major metabolites (betamethasone 17-propionate and MC180, respectively).

All available concentration results will be summarised by analyte and time point using appropriate descriptive statistics. Individual concentration versus time curves will be plotted (linear and semi-log plots) using actual time points.

Measured PK concentrations will be presented using standard descriptive statistics as described in section 7. Additionally, geometric mean and CV(%) will be presented.

Non-quantifiable (BLQ) levels of the analyte will be substituted by LLOQ for descriptive summaries and graphical presentation.

Plasma PK parameters at Week 4 (AUC<sub>0-t</sub>, AUC<sub>0-5</sub>, C<sub>max</sub>, and T<sub>max</sub>) will be calculated. The PK parameters AUC<sub>0-5</sub> and C<sub>max</sub> will be calculated using standard formulas inserting the LLOQ for non-quantifiable levels of the analyte. For a given analyte, the PK parameters AUC<sub>0-t</sub> and T<sub>max</sub> will be calculated if at least one post-dose time-point shows a quantifiable level of the analyte. PK parameter values will be rounded to the precision of the raw data from which it was derived (C<sub>max</sub>) or to 3 significant digits (AUC<sub>0-t</sub>, AUC<sub>0-5</sub>). T<sub>max</sub> will be rounded to two decimal places.

#### Pharmacokinetic Parameters Derivations:

**AUC**<sub>0-t</sub> (**pg\*h/mL**): The area under the curve spanning time interval from 0 to t (up to the last time point with measurable concentration above the quantification limit) will be calculated using the linear trapezoidal rule based on actual relative time of sampling.

- 1) Actual relative time of each sample will be derived as the difference between the datetime value of the corresponding sample and the datetime value of drug application, in hours. The time of the pre-dose sample will be set to 0.
- 2) For the calculation of AUC<sub>0-t</sub> BLQ values before the first reported measurable concentration (including pre-dose) will be substituted by LLOQ. The BLQ values after the last evaluable concentration will be set to missing.
- 3) Linear trapezoidal method is used. The area under the curve is defined as the sum of trapezoids across all pairs of time points from pre-dose to 5h post-dose at Visit 3 / Week 4.

#### Linear trapezoidal rule:

The area of the trapezoid between the two data points  $(t_1, C_1)$  and  $(t_2, C_2)$  where  $C_2 \ge C_1$  will be computed by:



 $AUC_{t1-t2}=0.5(t_2-t_1)(C_1+C_2).$ 

**AUC**<sub>0-5</sub> (**pg\*h/mL**): The area under the time-concentration curve from 0 to 5 hours will be calculated in a similar way to  $AUC_{0-t}$  (**pg\*h/mL**) while imputing the lower limit of quantification (LLoQ) for all concentrations below LLoQ.

C<sub>max</sub> (pg/mL): Individual Cmax values are directly determined from the plasma concentration time profiles of each subject as maximum of the observed concentration values after dosing. All BLQ values are substituted by LLOQ.

 $T_{max}$  (h): The time to attain  $C_{max}$ . If the same  $C_{max}$  concentration occurs at different time points,  $T_{max}$  is assigned to the first occurrence of  $C_{max}$ . If all concentrations are BLQ,  $T_{max}$  is not calculated.

The PK parameters will be summarised by analyte using standard descriptive statistics as described in section 7. Additionally, geometric mean and CV(%) will be presented for  $C_{max}$ ,  $AUC_{0-t}$  and  $AUC_{0-5}$ .

#### 11. Other Analyses

## 11.1. Physician global assessment

eCRF form: "PHYSICIAN'S GLOBAL ASSESSMENT OF PSORIASIS SEVERITY". Investigator ratings of disease severity (PGA) will be summarised by trial visit using frequency counts and percentages. The proportion of subjects with treatment success, defined as a minimum 2-point decrease from Baseline in the PGA on the trunk, limbs, and scalp will be summarised. Only subjects having at least moderate severity at baseline will be included in the summary of treatment success.

PGA results will be presented in accordance with section 7 by visit of assessment as scheduled in the Table 1 as the following outputs:

- descriptive statistics of measured values and changes from baseline by visit;
- number and proportion (95% CI) of subjects with treatment success, defined as a minimum
   2-point decrease from Baseline in the PGA;
- Shift table by post-baseline visit compared to baseline for PGA.

#### 11.2. Body surface area involvement

eCRF form: "BODY SURFACE AREA INVOLVEMENT ASSESSMENT".

The investigator or designee will assess the extent of the subject's psoriatic involvement on the scalp, neck, trunk and limbs (excluding face, genitals, and intertriginous areas).



The total psoriatic involvement on the scalp, neck, trunk and limbs will be recorded as a percentage of the total BSA, estimating that the surface of the subject's full, flat palm (including the five digits) correlates to approximately 1% of the total BSA.

Investigator assessment of BSA involvement for scalp and neck, trunk and/or limbs and total BSA involvement will be summarised in accordance with section 7 by visit of assessment as scheduled in the Table 1 as the following outputs:

descriptive statistics of BSA values and changes from baseline by visit.

#### 11.3. Psoriasis treatment convenience scale

eCRF form: "PSORIASIS TREATMENT CONVENIENCE SCALE".

The aim of PTCS is to assess the impact and convenience of psoriasis treatment. The scale consists of 6 disease-specific, self-reported questions with a recall period of 1 week and rated on a 1-10 scale.

- 1. How easy was the treatment to apply to the skin? Answered by 1 = very difficult to 10 = very easy.
- 2. How greasy was the treatment when applying it to the skin? Answered by 1 = very greasy to 10 = not greasy.
- 3. How moisturised did your skin feel after applying the treatment? Answered by 1 = not moisturized to 10 = very moisturized.
- 4. How greasy did your skin feel after applying the treatment? Answered by 1 = very greasy to 10 = not greasy.
- 5. How much did treating your skin disrupt your daily routine? Answered by 1 = very disturbing to 10 = not disturbing.
- 6. Overall, how satisfied were you with the medical treatment? Answered by 1 = not satisfied to 10 = very satisfied.

Ranging from 5 to 50, a PTCS total score is the sum of the scores on questions 1 to 5. If more than two questions are not answered, the PTCS total score is missing. If one or two questions remain unanswered, the missing scores are replaced by the average of the answered scores for the summation.

Psoriasis treatment convenience scale results will be presented by visit of assessment as scheduled in the Table 1.

Psoriasis treatment convenience scale results will be presented by visit as the following summaries:

- descriptive statistics for patient ratings by question;
- descriptive statistics for PTCS total score

All ratings will be listed.

#### 12. Reporting Conventions



Not Applicable.

#### 13. Technical Details

Statistical analysis will be performed using SAS 9.4.

Interim and final statistical analysis report will be prepared in the Microsoft Office Word (.docx) format. The results of statistical analysis will be presented in the form of tables, figures and listings in English.

#### 14. Summary of Changes to the Protocol

Due to small number of subjects at interim analysis geometric mean values of pharmacokinetic parameters will be directly derived from values of PK parameters calculated based on substitution of BLQ concentrations with LLOQ rather than estimated using parametric modelling. Median concentration – time plots will be omitted. Individual concentration – time plots will be presented instead.

#### 15. References

- 1) Committee for Proprietary Medicinal Products (CPMP). International Conference on Harmonisation (ICH) Topic E9: Note for Guidance on Statistical Principles for Clinical Trials; September 1998.
  - 2) DataMatrix SOP STAT001 Statistical Principles ver.3.0 June 2019.
- 3) DataMatrix\_SOP\_STAT002\_Statistical Analysis Plan Development\_ver.2.0\_July 2017.
- 4) DataMatrix\_SOP\_DM010\_Dictionary Management and Data Coding ver.2.0 August 2018.



#### 16. Listing of Tables, Listings and Figures

#### 16.1. Tables

- Table 14.1.1 Subject Disposition
- Table 14.1.2 Violation of Eligibility Criteria
- Table 14.1.4 Study Visits
- Table 14.1.5.1 Protocol Deviations
- Table 14.1.5.2 Major Protocol Deviations
- Table 14.1.6 Demographic Characteristics
- Table 14.1.7 Other Baseline Characteristics
- Table 14.1.8 Baseline Characteristics by Visit
- Table 14.1.9 Prior Medical Conditions/Diagnoses
- Table 14.1.10 Concurrent Medical Conditions/Diagnoses
- Table 14.1.11 Prior Therapy
- Table 14.1.12 Concomitant Therapy
- Table 14.1.13.1 Summary of Exposure and Compliance
- Table 14.1.13.2 Summary of Exposure and Compliance up to Week 2
- Table 14.1.13.3 Summary of Exposure and Compliance up to Week 4
- Table 14.1.13.4 Summary of Exposure and Compliance from Week 4 to Week 8
- Table 14.2.1.1 Individual and Summarized BDP Plasma Concentrations
- Table 14.2.1.2 Individual and Summarized Betamethasone 17-propionate Plasma Concentrations
- Table 14.2.1.3 Individual and Summarized CAL Plasma Concentrations
- Table 14.2.1.4 Individual and Summarized MC1080 Plasma Concentrations
- Table 14.2.2 Summary of Pharmacokinetic Parameters
- Table 14.3.1.1 Overall Summary of TEAEs
- Table 14.3.1.2.1 Incidence of Treatment-emergent Adverse Events
- Table 14.3.1.2.2 Incidence of Treatment-emergent Adverse Events up to Week 4
- Table 14.3.1.3.1 Incidence of Treatment-emergent Adverse Events Related to the Study Drug
- Table 14.3.1.3.2 Incidence of Treatment-emergent Adverse Events Related to the Study Drug up to Week 4
- Table 14.3.1.4.1 Incidence of Serious Treatment-emergent Adverse Events
- Table 14.3.1.4.2 Incidence of Serious Treatment-emergent Adverse Events up to Week 4
- Table 14.3.1.5.1 Incidence of Serious Treatment-emergent Adverse Events Related to the Study Drug
- Table 14.3.1.5.2 Incidence of Serious Treatment-emergent Adverse Events Related to the Study Drug up to Week 4
- Table 14.3.1.6.1 Incidence of Treatment-emergent Adverse Events by Maximum Severity
- Table 14.3.1.6.2 Incidence of Treatment-emergent Adverse Events up to Week 4 by Maximum Severity
- Table 14.3.1.7.1 Incidence of Treatment-Emergent Adverse Events by Closest Relationship
- Table 14.3.1.7.2 Incidence of Treatment-Emergent Adverse Events up to Week 4 by Closest Relationship
- Table 14.3.1.8.1 Incidence of Treatment-emergent Adverse Events Leading to Discontinuation of Study Drug
- Table 14.3.1.8.2 Incidence of Treatment-emergent Adverse Events Leading to Discontinuation of Study Drug up to Week 4
- Table 14.3.1.9.1 Incidence of Treatment-emergent Adverse Events Leading to Withdrawal



Table 14.3.1.9.2 Incidence of Treatment-emergent Adverse Events Leading to Withdrawal up to Week 4

Table 14.3.1.10.1 Incidence of Non-serious treatment-emergent Adverse Events Occurred at a Frequency of >=5%

Table 14.3.1.10.2 Incidence of Non-serious treatment-emergent Adverse Events Occurred at a Frequency of >=5% up to Week 4

Table 14.3.1.11 Incidence of Treatment-emergent Adverse Events Related to Cosyntropin

Table 14.3.1.12 Incidence of Treatment-emergent Adverse Events Related to Study Procedures

Table 14.3.2.1 Incidence of Treatment-emergent Adverse Events Leading to Death

Table 14.3.2.2 Incidence of Treatment-emergent Adverse Events Related to the Study Drug and Leading to Death

Table 14.3.4.1.1 Summary of ACTH Challenge Test

Table 14.3.4.1.2 Incidence of HPA Axis Suppression

Table 14.3.4.2.1 Summary of Calcium Metabolism Evaluation

Table 14.3.4.3.1 Summary of Hematology Parameters

Table 14.3.4.3.2 Summary of Blood Chemistry Parameters

Table 14.3.4.3.3 Summary of Morning Urine Assessment Parameters

Table 14.3.4.4.1 Hematology Shifts from Baseline

Table 14.3.4.4.2 Blood Chemistry Shifts from Baseline

Table 14.3.4.4.3 Morning Urine Assessment Shifts from Baseline

Table 14.3.4.5.1 Incidence of Hematology Assessments Outside of Normal Range

Table 14.3.4.5.2 Incidence of Blood Chemistry Assessments Outside of Normal Range

Table 14.3.4.5.3 Incidence of Morning Urine Assessments Outside of Normal Range

Table 14.3.4.6.1 Summary of Local Skin Reactions Assessment

Table 14.3.4.6.2 Local Skin Reactions Assessment Shifts from Baseline

Table 14.3.4.6.3 Summary of LSR Sum Score

Table 14.3.4.7.1 Summary of Vital Signs

Table 14.3.4.7.2 Incidence of Vital Signs Assessments Outside of Normal Range

Table 14.3.4.7.3 Incidence of Notably Abnormal Vital Signs Assessments

Table 14.3.4.8 Summary of Physical Parameters

Table 14.3.4.9 Summary of Physical Examination

Table 14.3.4.10.1 Summary of Electrocardiogram

Table 14.3.4.10.2 Incidence of Abnormal ECG Assessments

Table 14.3.4.10.3 Incidence of Notably Abnormal ECG Assessments

Table 14.4.1.1 Summary of PGA

Table 14.4.1.2 Summary of Treatment Success

Table 14.4.1.3 PGA Shifts from Baseline

Table 14.4.2.1 Summary of Body Surface Area Involvement

Table 14.4.3.1 Summary of Psoriasis Treatment Convenience Scale

#### 16.2. Figures

Figure 16.2.5.4 Individual BDP Plasma Concentration-time Profiles on Linear and Semilogarithmic Scales Week 4

Figure 16.2.5.5 Individual Calcipotriol (CAL) Plasma Concentration-time Profiles on Linear and Semi-logarithmic Scales Week 4



Figure 16.2.5.6 individual MC1080 Plasma Concentration-time Profiles on Linear and Semilogarithmic Scales Week 4

Figure 16.2.5.7 individual Betamethasone 17-propionate, Plasma Concentration-time Profiles on Linear and Semi-logarithmic Scales Week 4

#### 16.3. Listings

- Listing 16.2.1.1 Analysis Populations
- Listing 16.2.1.2 Subject Visits
- Listing 16.2.1.3 Study Completion
- Listing 16.2.1.4 Study Treatment Completion
- Listing 16.2.2.1 Violation of Inclusion/Exclusion Criteria
- Listing 16.2.2.2 Protocol Deviations
- Listing 16.2.4.1 Demographics and Other Baseline Characteristics
- Listing 16.2.4.2 Baseline Variables
- Listing 16.2.4.3 Medical History
- Listing 16.2.4.4 Prior/Concomitant Therapy
- Listing 16.2.4.5 Prior/Concomitant Procedures
- Listing 16.2.5.1 Exposure
- Listing 16.2.5.2 Study Drug Compliance
- Listing 16.2.5.3 Missed Doses
- Listing 16.2.5.4 Study Drug Accountability
- Listing 16.2.7.1 Adverse Events
- Listing 16.2.7.2 Serious Adverse Events
- Listing 16.2.7.3 Listing of Adverse Events Leading Discontinuation of Study Drug
- Listing 16.2.7.4 Listing of Adverse Events Leading to Withdrawal
- Listing 16.2.8.1 Hematology in SI Units
- Listing 16.2.8.2 Serum Biochemistry in SI Units
- Listing 16.2.8.3 Morning Urine Assessment in SI Units
- Listing 16.2.8.4 24-hour Urine Assessment
- Listing 16.2.8.5 Serum Pregnancy Test
- Listing 16.2.8.6 Urine Pregnancy Test
- Listing 16.2.8.7 ACTH Challenge Test
- Listing 16.2.8.8 Clinically Significant Laboratory Abnormalities
- Listing 16.2.9.1 Food Diary. Calcium-rich Nutrients Consumption
- Listing 16.2.9.2 Local Skin Reactions Assessment
- Listing 16.2.9.3 Vital Signs
- Listing 16.2.9.4 Electrocardiogram
- Listing 16.2.9.5 Physical Parameters
- Listing 16.2.9.6 Physical Examination
- Listing 16.2.9.7 Physician Global Assessment of Psoriasis Severity
- Listing 16.2.9.8 Body Surface Area Involvement
- Listing 16.2.9.9 Psoriasis Treatment Convenience Scale
- Listing 16.2.9.10 Pharmacokinetic Concentrations
- Listing 16.2.9.11 Pharmacokinetic Parameters



# MC2-01-C6\_STATISTICAL ANALYSIS PLAN\_Final 3.0\_07 September 2020 APPENDIX 1 TFLs Shells

# **Appendix 1. TFLs Shells**

**Tables Shells** 

**Subject Disposition** 

MC2 Therapeutics MC2-01-C6

#### Table 14.1.1 Subject Disposition

All Enrolled subjects
Page X of X

| | Total (N = XX) |
|---|---|
| | n (%) |
| Subjects who provided the informed consent / informed assent | XX |
| Screening Failures [1] | XX |
| Reasons for premature discontinuation | |
| Inconsistency with inclusion / exclusion criteria | XX |
| Withdrawal of informed consent / informed assent | XX |
| ••• | XX |
| Allocated to Treatment | XX |
| Safety Population | XX |
| HPA Population | XX (XX.X) |
| PK Population | XX (XX.X) |
| Completed the Study | XX (XX.X) |
| Discontinued the Study Prematurely | XX (XX.X) |
| Reasons for premature discontinuation | |
| Inconsistency with inclusion / exclusion criteria | XX (XX.X) |
| Lost to follow-up | XX (XX.X) |
| Withdrawal of informed consent / informed assent | XX (XX.X) |
| Intake of a prohibited medication(s) | XX (XX.X) |
| Pregnancy | XX (XX.X) |
| Adverse event / Serious adverse event | XX (XX.X) |
| Investigator's discretion | XX (XX.X) |
| Sponsor's decision to terminate the study | XX (XX.X) |


| Termination of the study by the Regulatory Authority | XX (XX.X) |
|---------------------------------------------------------------|-----------|
| Other | XX (XX.X) |
| Other reason 1 | XX (XX.X) |
| Other reason 2 | XX (XX.X) |
| ••• | XX (XX.X) |
| Discontinued Treatment before Week 8 visit | XX (XX.X) |
| Primary reason for treatment discontinuation | XX (XX.X) |
| Subject classified as clear at any of the on-treatment visits | XX (XX.X) |
| HPA axis suppression is noted at Week 4 | XX (XX.X) |
| Premature study termination | XX (XX.X) |
| Adverse event / Serious adverse event | XX (XX.X) |
| Investigator's discretion | XX (XX.X) |
| Other | XX (XX.X) |
| Other reason 1 | XX (XX.X) |
| Other reason 2 | XX (XX.X) |
| | XX (XX.X) |

HPA=Hypothalamic-pituitary-adrenal; PK=Pharmacokinetics.

[1] Including subjects who satisfied inclusion/exclusion criteria but who were not allocated to treatment (no drug dispensed).

N: the number of subjects in the All Enrolled subjects set.

n: the number of subjects within a specific category. Percentages are calculated based on the number of subjects in the Safety population.

Safety population: all subjects who are enrolled in the trial and dispensed the trial medication at Visit 1/Day 0, excluding subjects who return all of the trial medication unused.

PK population: all subjects in the Safety population who have received the planned application of treatment at the Week 4 visit and have had at least one blood draw for PK assessment at Week 4.

HPA population: all subjects in the Safety population that show normal HPA function at SV2.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings/ Datasets used/ Referenced Data Listings



MC2 Therapeutics MC2-01-C6

#### Table 14.1.2 Violation of Eligibility Criteria

Screening Failures
Page X of X

| | Total |
|-----------------------------------------------------|----------|
| | (N = XX) |
| Subjects with any violation of eligibility criteria | n<br>XX |
| Subjects with any violation of inclusion criteria | XX |
| Inclusion criterion #1 | XX |
| Inclusion criterion #2 | XX |
| ••• | ••• |
| Subjects with any violation of exclusion criteria | XX |
| Exclusion criterion #1 | XX |
| Exclusion criterion #2 | XX |
| ••• | • • • |

Inclusion criterion #1: The parent(s), or legal guardian(s) (according to national law) have provided written informed consent following their receipt of verbal and written information about the trial.

N: the number of Screening Failures.

n: the number of subjects within a specific category.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

**Programming Note:** Report only the criteria violated. If no criteria are violated suppress the printing of subsequent rows. Include description of all the criteria violated in the footnote.



MC2 Therapeutics

#### Table 14.1.4 Study Visits

Allocated to treatment set Page X of X

| | Total<br>(N = XX)<br>n (%) |
|------------------------------------|----------------------------|
| Screening Visit 1 (Days -42 to -8) | XX (XX.X) |
| Screening Visit 2 (Days -7 to -4) | XX (XX.X) |
| Visit 1 (Day 0) | XX (XX.X) |
| Visit 2 / Week 2 (Day 14 +/- 2) | XX (XX.X) |
| Visit 3 / Week 4 (Day 28 +/- 2) | XX (XX.X) |
| Visit 4 / Week 6 (Day 42 +/- 2) | XX (XX.X) |
| Visit 5 / Week 8 (Day 56 +/- 2) | XX (XX.X) |
| Follow-up Visit [1] | XX (XX.X) |
| Early Termination Visit | XX (XX.X) |

<sup>[1]</sup> Follow-up visit is required 2 weeks after the Week 8 visit. For subject with HPA axis suppression at Week 8 the follow-up visit should be 4 weeks after the Week 8 visit.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

N: the number of subjects in the Allocated to treatment set.

n: the number of subjects within a specific category. Percentages are calculated as (100 x n/N).



#### **Protocol Deviations**

MC2 Therapeutics MC2-01-C6

#### Table 14.1.5.1 Protocol Deviations

Allocated to treatment set Page X of X

| | Total<br>(N = XX)<br>n (%) |
|-----------------------------------------------|----------------------------|
| Subjects with at least one protocol deviation | XX (XX.X) |
| Deviation category #1 | XX (XX.X) |
| Deviation subcategory #1 | XX (XX.X) |
| Deviation subcategory #2 | XX (XX.X) |
| *** | |
| Deviation category #2 | XX (XX.X) |
| Deviation subcategory #1 | XX (XX.X) |
| Deviation subcategory #2 | XX (XX.X) |
| ••• | |

N: the number of subjects in the Allocated to treatment set.

n: the number of subjects with at least one protocol deviation. Percentages are calculated as (100 x n/N).

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

Similar to table 14.1.5.1, the following tables will be constructed (with corrections of underlined fragments in the footnote: "n: the number of subjects with at least one major protocol deviation."

Table 14.1.5.2 Major Protocol Deviations



### **Demographic Characteristics**

MC2 Therapeutics MC2-01-C6

#### Table 14.1.6 Demographic Characteristics

Safety population Page X of X

| | | Total (N = XX) |
|-------------------------------------------|-------|----------------|
| Country | | |
| n | | XX |
| Czech Republic | n (응) | XX (XX.X) |
| Germany | n (%) | XX (XX.X) |
| Hungary | n (%) | XX (XX.X) |
| Age (full years) | | |
| n | | XX |
| Mean | | XX.X |
| SD | | XX.X |
| Median | | XX.X |
| Q1, Q3 | | XX.X, XX.X |
| Min, Max | | XX.X, XX.X |
| Sex | | |
| n | | XX |
| Male | n (응) | XX (XX.X) |
| Female | n (%) | XX (XX.X) |
| Unknown | n (%) | XX (XX.X) |
| thnic origin | | |
| n | | XX |
| Hispanic or Latino | n (%) | XX (XX.X) |
| Not Hispanic or Latino | n (%) | XX (XX.X) |
| Unknown | n (%) | XX (XX.X) |
| Race | | |
| n | | XX |
| American Indian or Alaska Native | n (%) | XX (XX.X) |
| Asian | n (%) | XX (XX.X) |
| Black or African American | n (%) | XX (XX.X) |
| Native Hawaiian or Other Pacific Islander | | |



| White<br>Other / Multiple | n (%) | XX (XX.X) |
|---------------------------|-------|-----------|
| Other race 1 | n (%) | XX (XX.X) |
| Other race 2 | n (%) | xx (xx.x) |
| ••• | ••• | |
| Unknown | n (%) | XX (XX.X) |

N: the number of subjects in the Safety population.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

n: the number of valid measurements or the number of subjects within a specific category. Percentages are calculated as  $(100 \times n/N)$ .



#### **Baseline Variables**

MC2 Therapeutics MC2-01-C6

#### Table 14.1.7 Other Baseline Characteristics

Safety population Page X of X

| | Total<br>(N = XX) |
|-------|-------------------------------------|
| | XX |
| n (%) | XX (XX.X) |
| n (%) | XX (XX.X) |
| n (%) | XX (XX.X) |
| n (%) | XX (XX.X) |
| n (%) | XX (XX.X) |
| n (%) | XX (XX.X) |
| n (%) | XX (XX.X) |
| • • • | • • • |
| | n (%) n (%) n (%) n (%) n (%) n (%) |

N: the number of subjects in the Safety population.

n: the number of valid measurements or the number of subjects within a specific category. Percentages are calculated as  $(100 \times n/N)$ . Duration of disease is calculated in months as (date of diagnosis - date of informed consent + 1) / 30.4375.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming Note:** Continue table for the following parameters:

- Duration of disease (months) (Continuous);
- Previous treatment (Biologics and systemic [TNF-a inhibitors, IL-12/23 inhibitors, IL-17 inhibitors, Fumarate, Other], Phototherapy (UVA or PUVA), Topical: fixed combination corticosteroid plus vitamin D analogs, Topical: corticosteroids, Topical: retinoids, Topical: salicylic acid, Topical: vitamin D analogs, Topical: calcineurin inhibitors, Topical: tar, Other).



MC2 Therapeutics MC2-01-C6

#### Table 14.1.8 Baseline Characteristics by Visit

Safety population

Page X of X

Parameter: Physician global assessment of psoriasis severity (categorical)

| | Total |
|------------------|-----------|
| Visit | (N = XX) |
| | n (%) |
| Screening V1 | |
| | XX |
| n<br>O - Clear | |
| 1 - Almost Clear | XX (XX.X) |
| 2 - Mild | XX (XX.X) |
| | XX (XX.X) |
| 3 - Moderate | XX (XX.X) |
| 4 - Severe | XX (XX.X) |
| Screening V2 | |
| n | xx |
| 0 - Clear | XX (XX.X) |
| 1 - Almost Clear | XX (XX.X) |
| 2 - Mild | XX (XX.X) |
| 3 - Moderate | XX (XX.X) |
| 4 - Severe | XX (XX.X) |
| Visit 1 (Day 0) | |
| n | XX |
| 0 - Clear | XX (XX.X) |
| 1 - Almost Clear | XX (XX.X) |
| 2 - Mild | XX (XX.X) |
| 3 - Moderate | XX (XX.X) |
| 4 - Severe | XX (XX.X) |
| Baseline [1] | |
| n | XX |
| 0 - Clear | XX (XX.X) |
| 1 - Almost Clear | XX (XX.X) |
| 2 - Mild | XX (XX.X) |
| 3 - Moderate | XX (XX.X) |
| 4 - Severe | |
| A - Severe | XX (XX.X) |



BMI=Body Mass Index; BSA=Body Surface Area; PGA= Physician Global Assessment.

N: the number of subjects in the Safety population.

n: the number of subjects within a specific category or the number of valid observations. Percentages are based on the corresponding number of valid observations.

[1] Baseline is the last non-missing assessment prior to the first dose of the study drug.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

#### **Programming note:**

Report the following visits: Screening V1, Screening V2, Visit 1 (Day 0), Baseline (where applicable). Continue table for the following parameters:

- Physician global assessment of psoriasis severity (continuous);
- Height (cm);
- Weight (kg);
- Body mass index (BMI, kg/m2);
- Systolic blood pressure (mm Hg);
- Diastolic blood pressure (mm Hg);
- Pulse (beats/min);
- Oral temperature (C);
- Tympanic temperature (C);
- 25-Hydroxyvitamin D3 (ug/L);
- Serum Calcium Corrected for Albumin (mmol/L);
- Scalp BSA psoriatic involvement (%);
- Neck, Trunk and/or Limbs BSA psoriatic involvement (%);
- Total psoriatic involvement (%);
- Serum cortisol pre-stimulation (nmol/L);
- Serum cortisol post-stimulation (nmol/L);
- Investigator assessment of Erosion/ulceration in lesional area (0 (Absent), 1 (Mild), 2 (Moderate), 3 (Severe));
- Investigator assessment of Vesicles in lesional area (0 (Absent), 1 (Mild), 2 (Moderate), 3 (Severe));
- Investigator assessment of Erythema in perilesional area (0 (Absent), 1 (Mild), 2 (Moderate), 3 (Severe));



- Investigator assessment of Scaling in the perilesional area (0 (Absent), 1 (Mild), 2 (Moderate), 3 (Severe));
- Investigator assessment of Edema in perilesional area (0 (Absent), 1 (Mild), 2 (Moderate), 3 (Severe));
- Investigator assessment of Atrophy in perilesional area (0 (Absent), 1 (Mild), 2 (Moderate), 3 (Severe));
- Investigator assessment of Vesicles in perilesional area (0 (Absent), 1 (Mild), 2 (Moderate), 3 (Severe));
- Investigator assessment of Erosion/ulceration in perilesional area (0 (Absent), 1 (Mild), 2 (Moderate), 3 (Severe)).



### **Medical History**

MC2 Therapeutics

#### Table 14.1.9 Prior Medical Conditions/Diagnoses

Safety population Page X of X

| System Organ Class (SOC) Preferred Term (PT) | Total<br>(N = XX) |
|----------------------------------------------|-------------------|
| | n (%) |
| Overall | XX (XX.X) |
| System Organ Class 1 | XX (XX.X) |
| Preferred Term 1 | XX (XX.X) |
| Preferred Term 2 | XX (XX.X) |
| • • • | ••• |
| System Organ Class 2 | XX (XX.X) |
| Preferred Term 1 | XX (XX.X) |
| Preferred Term 2 | XX (XX.X) |
| ••• | ••• |
| ••• | • • • |

MedDRA=Medical Dictionary for Regulatory Activities.

N: the number of subjects in the Safety population.

n: the number of subjects with at least one medical history event within a specific category. Percentages are calculated as  $(100 \times n/N)$ . Conditions/diagnoses are classified as 'Prior' if the condition/diagnosis end date is prior to study treatment start date or the subject did not receive any study treatment.

Medical history events are coded using MedDRA version XX.X.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

**Programming note:** System organ classes (SOC) and preferred terms (PT) within each SOC are sorted in descending order of n(%).



Similar to table 14.1.9, the following table will be constructed (with corrections of underlined footnote: "Conditions/diagnoses are classified as 'Concurrent' if the condition/diagnosis end date is on or after the study treatment start date") for the Safety population:

Table 14.1.10 Concurrent Medical Conditions/Diagnoses



### **Prior and Concomitant therapy**

MC2 Therapeutics
MC2-01-C6

Table 14.1.11 Prior Therapy
Safety population
Page X of X

| Pharmacological subgroup (3rd level) | Total |
|--------------------------------------|----------------|
| Chemical substance (5th level) | (N = XX) n (%) |
| Overall | XX (XX.X) |
| Pharmacological subgroup 1 | XX (XX.X) |
| Chemical substance 1 | XX (XX.X) |
| Chemical substance 2 | XX (XX.X) |
| • • • | |
| Pharmacological subgroup 2 | XX (XX.X) |
| Chemical substance 1 | XX (XX.X) |
| Chemical substance 2 | XX (XX.X) |
| ••• | |
| | • • • |

N: the number of subjects in the Safety population.

Medications are coded by WHO drug dictionary version XX.X.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

**Programming note:** The pharmacological subgroups and chemical substances within each pharmacological subgroup are sorted in descending order of n (%). Each subject is counted only once per pharmacological subgroup and once per chemical substance.

n: the number of subjects with at least one  $\underline{\text{prior}}$  medication within a specific category. Percentages are calculated as (100 x n/N). Medications are classed as 'Prior' if the medication end date is prior to study treatment start date or the subject did not receive any study treatment.



Similar to table 14.1.11, the following table will be constructed (with corrections of underlined fragments in the footnote: "Medication is classified as 'Concomitant' if either the medication start date is on or after study treatment start date and on or prior to study treatment end date, or the medication start date is before the study treatment end date and the medication end date is on or after the study treatment start date." for the Safety population:

Table 14.1.12 Concomitant Therapy





**Exposure** 

MC2 Therapeutics MC2-01-C6

#### Table 14.1.13.1 Summary of Exposure and Compliance

Safety population Page X of X

| | | $ \text{Total} \\ (N = XX) $ |
|---|---|---|
| otal duration of exposure (days) | | |
| n | | XX |
| Mean | | XX.X |
| SD | | XX.X |
| Median | | XX.X |
| Q1, Q3 | | XX.X, XX.X |
| Min, Max | | XX, XX |
| | | · |
| xtent of exposure (days) | | |
| n<br> | | XX |
| Mean | | XX.X |
| SD | | XX.X |
| Median | | XX.X |
| Q1, Q3 | | XX.X, XX.X |
| Min, Max | | XX, XX |
| ompliance (%) | | |
| n | | XX |
| Mean | | XX.XX |
| SD | | XX.XX |
| Median | | XX.XX |
| Q1, Q3 | | XX.XX, XX.XX |
| Min, Max | | XX.X, XX.X |
| ompliance category | . (0) | 1717 (1717 17) |
| < 80% | n (%) | XX (XX.X) |
| >= 80% | n (%) | XX (XX.X) |
| verage weekly dose (g) | | |
| n | | XX |



| Mean<br>SD<br>Median<br>Q1, Q3<br>Min, Max | XX.XX<br>XX.XX<br>XX.XX<br>XX.XX, XX.XX<br>XX.X, XX.X |
|---|---|
| Total dose (g) | |
| n | XX |
| Mean | XX.XX |
| SD | XX.XX |
| Median | XX.XX |
| Q1, Q3 | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X |
| Number of missed doses (subjects with at least 1 missed dose) [1] | |
| n | XX |
| Mean | XX.X |
| SD | XX.X |
| Median | XX.X |
| Q1, Q3 | XX.X, XX.X |
| Min, Max | XX, XX |
| Number of missed doses (including zero counts) [2] | |
| n | XX |
| Mean | XX.X |
| SD | XX.X |
| Median | XX.X |
| Q1, Q3 | XX.X, XX.X |
| Min, Max | XX, XX |

N: the number of subjects in the Safety population.

n: the number of valid measurements or the number of subjects within a specific category. Percentages are calculated as  $(100 \times n/N)$ .

Total duration of exposure (days) is defined as (date of the last dose - date of the first dose + 1).

Total dose (g) is assessed as (weight of the tube dispensed - weight of the tube returned) summed over all tubes used and returned. Lost and unused tubes were not accounted for in the calculation of total dose.

Extent of exposure (days) is defined as (number of required days - number of missed doses).

Compliance is estimated as [100% \* (number of required days - number of missed doses) / number of required days].

Periods of approved discontinuations are not taken into account in the calculation of extent of exposure and compliance.

- [1] Only subjects with at least one missed dose were included into this summary.
- [2] Subjects with no missed doses during the period are included with zero counts.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings





Similar to table 14.1.13.1, the following tables will be constructed:

Table 14.1.13.2 Summary of Exposure and Compliance up to Week 2
Table 14.1.13.3 Summary of Exposure and Compliance up to Week 4
Table 14.1.13.4 Summary of Exposure and Compliance from Week 4 to Week 8



### **Pharmacokinetics Analyses**

MC2 Therapeutics MC2-01-C6

#### Table 14.2.1.1 Individual and Summarized BDP Plasma Concentrations

PK population Page X of X

| Subject Number/<br>Statistic | SV2 | Week 2<br>pre-dose | Week 4<br>pre-dose | 1h | 3h | 5h | Week 8<br>pre-dose |
|---|---|---|---|---|---|---|---|
| xxxxxxxxxxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| XXXXXXXXXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| XXXXXXXXXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| XXXXXXXXXXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| xxxxxxxxxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| n | XX | XX | XX | XX | XX | XX | XX |
| nquant | XX | XX | XX | XX | XX | XX | XX |
| Mean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| gMean | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| gCV (%) | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.XX | XX.X, XX.XX | XX.X, XX.XX | XX.X, XX.XX | XX.X, XX.XX | XX.X, XX.XX | XX.X, XX.X |
| Min, Max | XX.XX, XX.X | XX.XX, XX.X | XX.XX, XX.X | XX.XX, XX.X | XX.XX, XX.X | XX.XX, XX.X | XX.XX, XX. |

BDP=Betamethasone dipropionate; BLQ=Below Limit of Quantification; gCV=Geometric Coefficient of Variation; gMean=Geometric Mean; LLOQ=Lower Limit of Quantification; PK=Pharmacokinetic.

BLQ concentrations were substituted with LLOQ for the calculation of summary statistics. LLOQ for  $\underline{BDP}$  is XX.X  $\underline{pg/mL}$ .

The unit of concentration is pg/mL.

n: the number of valid measurements; nquant: number of measurements with quantifiable level of analyte.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

Similar to table 14.2.1.1, the following tables will be constructed (with modification of underlined fragments):





Table 14.2.1.2 Individual and Summarized Betamethasone 17-propionate Plasma Concentrations

Table 14.2.1.3 Individual and Summarized CAL Plasma Concentrations

Table 14.2.1.4 Individual and Summarized MC1080 Plasma Concentrations

#### **Programming note:**

Change the corresponding footnote to "CAL=Calcipotriene (Calcipotriol)".





MC2 Therapeutics MC2-01-C6

#### Table 14.2.2 Summary of Pharmacokinetic Parameters

PK population Page X of X

Analyte: Betamethasone dipropionate (BDP)

| Cmax (pg/mL) | |
|------------------|--------------|
| n | XX |
| Mean | XX.XX |
| SD | XX.XX |
| gMean | XX.XX |
| gCV(%) | XX.XX |
| Median | XX.XX |
| Q1, Q3 | XX.XX, XX.XX |
| Min, Max | XX.XX, XX.XX |
| AUCO-5 (pg*h/mL) | |
| n | XX |
| Mean | XX.XX |
| SD | XX.XX |
| gMean | XX.XX |
| gCV (%) | XX.X |
| Median | XX.XX |
| Q1, Q3 | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X |
| | MATAY MATA |
| UCO-t (pg*h/mL) | |
| n | XX |
| Mean | XX.XX |
| SD | XX.XX |
| gMean | XX.XX |
| gCV(%) | XX.X |
| Median | XX.XX |
| Q1, Q3 | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X |
| max (h) | |
| n | XX |
| Mean | XX.XX |
| SD | XX.XX |





AUC= Area under the time-concentration curve; BDP=Betamethasone dipropionate; CAL=Calcipotriene (Calcipotriol); Cmax= Maximum plasma drug concentration; gCV=Geometric Coefficient of Variation; gMean=Geometric Mean; PK=Pharmacokinetic; Tmax= Time to maximum plasma drug concentration.

N: the number of subjects in the PK population.

n: the number of valid measurements.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

#### **Programming note:**

Continue table for the following analytes:

- Betamethasone 17-propionate;
- Calcipotriene (Calcipotriol, CAL);
- MC1080.



### **Safety Analyses**

**Adverse Events** 

MC2 Therapeutics MC2-01-C6

#### Table 14.3.1.1 Overall Summary of TEAEs

Safety population Page X of X

| | Total |
|----------------------------------------------------|----------------|
| | (N = XX) |
| | n (%) / E |
| Any TEAE | XX (XX.X) / XX |
| any TEAE related to study treatment | XX (XX.X) / XX |
| ny TEAE related to study procedures | XX (XX.X) / XX |
| any TEAE related to Cosyntropin | XX (XX.X) / XX |
| any Serious TEAE | XX (XX.X) / XX |
| ny Serious TEAE related to study treatment | XX (XX.X) / XX |
| ny TEAE leading to study treatment discontinuation | XX (XX.X) / XX |
| any TEAE leading to withdrawal | XX (XX.X) / XX |
| aximum Severity | |
| Mild | XX (XX.X) |
| Moderate | XX (XX.X) |
| Severe | XX (XX.X) |
| trongest Causal Relationship to Study Treatment | |
| Not related | XX (XX.X) |
| Possibly related | XX (XX.X) |
| Probably related | XX (XX.X) |
| Definitely related | XX (XX.X) |

AE=Adverse Event; TEAE=Treatment-Emergent Adverse Event.

N: the number of subjects in the Safety population.

n: the number of subjects with at least one TEAE within a specific category. Percentages are calculated as  $(100 \times n/N)$ .

E: total number of TEAEs reported within a specific category.

A TEAE is defined as an AE that started after the first dose of the study treatment.

If the severity is missing for a TEAE, then 'Severe' category is assigned.

If the relationship is missing for a TEAE, then 'Definitely related' category is assigned.





Subjects with more than one TEAE will be counted once in the maximum severity or strongest relationship category.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings



MC2 Therapeutics MC2-01-C6

#### Table 14.3.1.2.1 Incidence of Treatment-emergent Adverse Events

Safety population Page X of X

| System Organ Class (SOC) | Total $(N = XX)$ |
|--------------------------|-----------------------|
| Preferred Term (PT) | (N - AA)<br>n (%) / E |
| Overall | XX (XX.X) / XX |
| System Organ Class 1 | XX (XX.X) / XX |
| Preferred Term 1 | XX (XX.X) / XX |
| Preferred Term 2 | XX (XX.X) / XX |
| System Organ Class 2 | XX (XX.X) / XX |
| Preferred Term 1 | XX (XX.X) / XX |
| Preferred Term 2 | XX (XX.X) / XX |
| ••• | |

AE=Adverse Event; MedDRA=Medical Dictionary for Regulatory Activities; TEAE=Treatment-Emergent Adverse Event.

N: the number of subjects in the Safety population.

n: the number of subjects with at least one TEAE within a specific category. Percentages are calculated as  $(100 \times n/N)$ .

 $\mathtt{E}\colon \mathtt{total}\ \mathtt{number}\ \mathtt{of}\ \underline{\mathtt{TEAEs}}\ \mathtt{reported}\ \mathtt{within}\ \mathtt{a}\ \mathtt{specific}\ \mathtt{category}.$ 

Adverse events are coded by MedDRA version XX.X.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

System organ classes (SOC) and preferred terms (PT) within each SOC should be sorted in descending order of n (%). Each subject is counted only once per preferred term (PT) and once per system organ class (SOC).



Similar to table 14.3.1.2.1, the following tables will be constructed (with the corresponding corrections of underlined fragments in the note):

```
Table 14.3.1.2.2 Incidence of Treatment-emergent Adverse Events up to Week 4
Table 14.3.1.3.1 Incidence of Treatment-emergent Adverse Events Related to the Study Drug
Table 14.3.1.3.2 Incidence of Treatment-emergent Adverse Events Related to the Study Drug up to Week 4
Table 14.3.1.4.1 Incidence of Serious Treatment-emergent Adverse Events
Table 14.3.1.4.2 Incidence of Serious Treatment-emergent Adverse Events up to Week 4
Table 14.3.1.5.1 Incidence of Serious Treatment-emergent Adverse Events Related to the Study Drug
Table 14.3.1.5.2 Incidence of Serious Treatment-emergent Adverse Events Related to the Study Drug up to Week 4
```



MC2 Therapeutics MC2-01-C6

#### Table 14.3.1.6.1 Incidence of Treatment-emergent Adverse Events by Maximum Severity

Safety population Page X of X

| System Organ Class (SOC) | | Total |
|--------------------------|----------|----------------|
| Preferred Term (PT) | Severity | (N = XX) |
| rielelled lelm (ri) | | n (%) / E |
| Overall | Mild | XX (XX.X) / XX |
| | Moderate | XX (XX.X) / XX |
| | Severe | XX (XX.X) / XX |
| System Organ Class 1 | Mild | XX (XX.X) / XX |
| | Moderate | XX (XX.X) / XX |
| | Severe | XX (XX.X) / XX |
| Preferred Term 1 | Mild | XX (XX.X) / XX |
| | Moderate | XX (XX.X) / XX |
| | Severe | XX (XX.X) / XX |
| Preferred Term 2 | Mild | XX (XX.X) / XX |
| | Moderate | XX (XX.X) / XX |
| | Severe | XX (XX.X) / XX |
| ••• | ••• | |
| System Organ Class 2 | Mild | XX (XX.X) / XX |
| | Moderate | XX (XX.X) / XX |
| | Severe | XX (XX.X) / XX |
| ••• | ••• | ••• |

AE=Adverse Event; MedDRA=Medical Dictionary for Regulatory Activities; TEAE=Treatment-Emergent Adverse Event.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

N: the number of subjects in the Safety population.

n: the number of subjects with at least one TEAE within a specific category. Percentages are calculated as  $(100 \times n/N)$ .

E: total number of TEAEs reported with appropriate severity.

For 'Overall' and for each SOC and SOC/PT, each subject is counted once in the category of the maximum severity.

For 'Overall', the number of all reported TEAEs are presented; for each SOC and SOC/PT, the number of TEAEs of maximum severity is given.

If the severity is missing for a TEAE, then 'Severe' category is assigned.

AEs are coded using MedDRA version XX.X.



### **Programming note:**

System organ classes (SOC) and preferred terms (PT) within each SOC should be sorted in descending order of n (%).

Similar to table 14.3.1.6.1, the following tables will be constructed:

Table 14.3.1.6.2 Incidence of Treatment-emergent Adverse Events up to Week 4 by Maximum Severity



MC2 Therapeutics MC2-01-C6

#### Table 14.3.1.7.1 Incidence of Treatment-Emergent Adverse Events by Closest Relationship

Safety population Page X of X

| System Organ Class (SOC) | | Total |
|--------------------------|--------------------|----------------|
| Preferred Term (PT) | Relationship | (N = XX) |
| rielelled leim (F1) | | n (%) / E |
| Overall | Not related | XX (XX.X) / XX |
| | Possibly related | XX (XX.X) / XX |
| | Probably related | XX (XX.X) / XX |
| | Definitely related | XX (XX.X) / XX |
| System Organ Class 1 | Not related | XX (XX.X) / XX |
| | Possibly related | XX (XX.X) / XX |
| | Probably related | XX (XX.X) / XX |
| | Definitely related | XX (XX.X) / XX |
| Preferred Term 1 | Not related | XX (XX.X) / XX |
| | Possibly related | XX (XX.X) / XX |
| | Probably related | XX (XX.X) / XX |
| | Definitely related | XX (XX.X) / XX |
| Preferred Term 2 | Not related | XX (XX.X) / XX |
| | Possibly related | XX (XX.X) / XX |
| | Probably related | XX (XX.X) / XX |
| | Definitely related | XX (XX.X) / XX |
| System Organ Class 2 | Not related | XX (XX.X) / XX |
| -<br>- | Possibly related | XX (XX.X) / XX |
| | Probably related | XX (XX.X) / XX |
| | Definitely related | XX (XX.X) / XX |
| | ••• | |

AE=Adverse Event; MedDRA=Medical Dictionary for Regulatory Activities; TEAE=Treatment-Emergent Adverse Event.

N: the number of subjects in the Safety population.

n: the number of subjects with at least one TEAE within a specific category. Percentages are calculated as  $(100 \times n/N)$ .

E: total number of TEAEs reported with given category of relationship to study drug.

For 'Overall' and for each SOC and SOC/PT, each subject is counted once in the category of the closest relationship.

For 'Overall', the number of all reported TEAEs are presented; for each SOC and SOC/PT, the number of TEAEs of closest relationship is given.



If the relationship is missing for a TEAE, then 'Definitely related' category is assigned. AEs are coded using MedDRA version XX.X.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

#### **Programming note:**

System organ classes (SOC) and preferred terms (PT) within each SOC should be sorted in descending order of n (%).

Similar to table 14.3.1.7.1, the following tables will be constructed (with the corresponding corrections of underlined fragments in the note):

Table 14.3.1.7.2 Incidence of Treatment-Emergent Adverse Events up to Week 4 by Closest Relationship

Similar to table 14.3.1.2.1, the following tables will be constructed (with the corresponding corrections of underlined fragments in the note):

Table 14.3.1.8.1 Incidence of Treatment-emergent Adverse Events Leading to Discontinuation of Study Drug up to Week 4
Table 14.3.1.8.2 Incidence of Treatment-emergent Adverse Events Leading to Withdrawal
Table 14.3.1.9.1 Incidence of Treatment-emergent Adverse Events Leading to Withdrawal
Table 14.3.1.9.2 Incidence of Treatment-emergent Adverse Events Leading to Withdrawal up to Week 4
Table 14.3.1.10.1 Incidence of Non-serious treatment-emergent Adverse Events Occurred at a Frequency of >=5%
Table 14.3.1.10.2 Incidence of Non-serious treatment-emergent Adverse Events Occurred at a Frequency of >=5% up to Week 4
Table 14.3.1.11 Incidence of Treatment-emergent Adverse Events Related to Cosyntropin
Table 14.3.1.12 Incidence of Treatment-emergent Adverse Events Related to Study Procedures
Table 14.3.2.1 Incidence of Treatment-emergent Adverse Events Leading to Death
Table 14.3.2.2 Incidence of Treatment-emergent Adverse Events Related to the Study Drug and Leading to Death



### **HPA Axis Suppression**

MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.1.1 Summary of ACTH Challenge Test

HPA population Page X of X

| Serum Cortisol (nmol/L) | Total<br>(N=XX) | |
|-------------------------|-----------------------|-----------------------|
| | Pre-stimulation | Post-stimulation |
| Baseline | | |
| n | XX | XX |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | XX.XX [XX.XX - XX.XX] |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |
| Visit 3 / Week 4 | | |
| n | XX | XX |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | XX.XX [XX.XX - XX.XX] |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |
| Visit 5 / Week 8 | | |
| n | XX | XX |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | XX.XX [XX.XX - XX.XX] |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |
| Follow-up | | |
| n | XX | XX |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | XX.XX [XX.XX - XX.XX] |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |





HPA=Hypothalamic-pituitary-adrenal.

N: the number of subjects in the HPA population. n: the number of valid measurements.

Measurements of serum cortisol levels pre- and post- stimulation with cosyntropin 0.25 mg are presented.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings



MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.1.2 Incidence of HPA Axis Suppression

HPA population Page X of X

| | | Total (N = XX) |
|---|---|---|
| HPA axis suppression | | |
| Overall | n' (%) [1]<br>n (%) [2]<br>95% CI | XX (XX.X)<br>XX (XX.X)<br>XX.X, XX.X |
| Visit 3 / Week 4 | n' (%) [1]<br>n (%) [2]<br>95% CI | XX (XX.X)<br>XX (XX.X)<br>XX.X, XX.X |
| Visit 5 / Week 8 | n' (%) [1]<br>n (%) [2]<br>95% CI | XX (XX.X)<br>XX (XX.X)<br>XX.X, XX.X |
| HPA axis suppressed at Week 4 | n' (%) [3]<br>n (%) [2]<br>95% CI | XX (XX.X)<br>XX (XX.X)<br>XX.X, XX.X |
| HPA axis not suppressed at Week 4 | n' (%) [3]<br>n (%) [2]<br>95% CI | XX (XX.X)<br>XX (XX.X)<br>XX.X, XX.X |

CI=Confidence Interval; HPA=Hypothalamic-pituitary-adrenal.

Confidence interval is calculated using Clopper-Pearson method.

Adrenal suppression is defined as the 30-minute post-stimulation serum cortisol level below 18 ug/dL (500 nmol/L).

N: the number of subjects in the HPA population. n: the number of subjects within a specific category. n': the number of valid observations.

<sup>[1]</sup> Subjects having any post-baseline values (for 'Overall' category) or values at the corresponding visit. Percentage is calculated as (100 x n/N).

<sup>[2]</sup> Percentages are based on the corresponding number of valid observations.

<sup>[3]</sup> Subjects with corresponding HPA suppression status at Week 4 having values at Visit 5 / Week 8. Percentage is calculated based on number of subjects with corresponding HPA suppression status at Week 4.





Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings



#### **Calcium Metabolism**

MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.2.1 Summary of Calcium Metabolism Evaluation

Safety population Page X of X

Parameter: Serum Calcium Corrected for Albumin (mmol/L)

| | Total (N = XX) | Change from the baseline |
|------------------|-----------------------|--------------------------|
| Baseline | | |
| n | XX | |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | |
| SD | XX.XX | |
| Median | XX.XX | |
| Q1, Q3 | XX.XX, XX.XX | |
| Min, Max | XX.X, XX.X | |
| Visit 3 / Week 4 | | |
| n | XX | XX |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | XX.XX [XX.XX - XX.XX] |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |
| Visit 5 / Week 8 | | |
| n | XX | XX |
| Mean [95% CI] | XX.XX [XX.XX - XX.XX] | XX.XX [XX.XX - XX.XX] |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |

N: the number of subjects in the Safety population. n: the number of valid measurements.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**





Report the following parameters: Serum Calcium (mmol/L), Urinary Calcium/Creatinine (mmol/mmol).



### **Clinical Laboratory Evaluation**

MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.3.1 Summary of Hematology Parameters

Safety population Page X of X

Parameter: XXXXXXXXXXXXXXXX (units)

| | Total (N = XX) | Change from the baseline |
|-----------------------|----------------|--------------------------|
| Paraller. | | |
| Baseline | 777 | |
| n<br>Wasan | XX | |
| Mean | XX.XX | |
| SD | XX.XX | |
| Median | XX.XX | |
| Q1, Q3 | XX.XX, XX.XX | |
| Min, Max | XX.X, XX.X | |
| Visit 3 / Week 4 | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |
| Visit 5 / Week 8 | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |
| Highest post-baseline | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |


| n | XX | XX |
|----------|--------------|--------------|
| Mean | XX.XX | XX.XX |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |

N: the number of subjects in the Safety population.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug application.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Report the following parameters: Hemoglobin (mmol/L), Hematocrit (L/L), Erythrocytes (10^12/L), MCV (fL), Leukocytes (10^9/L), Lymphocytes (10^9/L), Lymphocytes (%), Monocytes (%), Monocytes (%), Neutrophils (10^9/L), Neutrophils (10^9/L), Neutrophils (10^9/L), Basophils (10^9/L), Eosinophils (10^9/L), Eosinophils (10^9/L).

Similar to table 14.3.4.3.1, the following tables will be constructed:

#### Table 14.3.4.3.2 Summary of Blood Chemistry Parameters

Report the following parameters: Urea (mmol/L), Urea Nitrogen (mmol/L), Serum Glucose (mmol/L), Serum Creatinine (umol/L), Serum Albumin (g/L), Sodium (mmol/L), Potassium (mmol/L), Chloride (mmol/L), Serum Phosphate (mmol/L), Alkaline Phosphatase (U/L), Parathyroid Hormone (pmol/L).

#### Table 14.3.4.3.3 Summary of Morning Urine Assessment Parameters

Report the following parameters: Urinary Calcium (mmol/L), Total Calcium Excretion (mmol), Urinary Phosphate (mmol/L), Total Phosphate Excretion (mmol), Urinary Creatinine (g/L), Total Creatinine Excretion (g), Urinary Phosphate/Creatinine (mg/g), Volume (mL).

n: the number of valid measurements.



MC2 Therapeutics MC2-01-C6

### Table 14.3.4.4.1 Hematology Shifts from Baseline

Safety population Page X of X

Parameter: XXXXXXXXXXXXXXX (units)

| | _ | Baseline | | | |
|---|---|---|---|---|---|
| | | Low | Normal | High | Total |
| Visit 3 / Week 4 | | | | | |
| Low | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Visit 5 / Week 8 | | | | | |
| Low | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Highest post-baseline | | | | | |
| Low | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Lowest post-baseline | | | | | |
| Low | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Normal | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| High | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |

The baseline value for a variable is defined as the last non-missing value collected before the first study drug application.

Percentages are based on the number of subjects with non-missing assessment at the corresponding time point and at baseline.

For highest/lowest post-baseline values percentages are based on the number of subjects with non-missing assessment at baseline and at least one non-missing post-baseline assessment for the corresponding parameter.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings





Similar to table 14.4.2.2.1, the following tables will be constructed:

Table 14.3.4.4.2 Blood Chemistry Shifts from Baseline Table 14.3.4.4.3 Morning Urine Assessment Shifts from Baseline



MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.5.1 Incidence of Hematology Assessments Outside of Normal Range

Safety population Page X of X

Parameter: XXXXXXXXXXXXXXX (units)

| | Total |
|------------------|-----------|
| | (N = XX) |
| | n (%) |
| verall | |
| n [1] | XX |
| Out of Range | XX (XX.X) |
| Low | XX (XX.X) |
| High | XX (XX.X) |
| saseline | |
| n | XX |
| Normal | XX (XX.X) |
| Out of Range | XX (XX.X) |
| Low | XX (XX.X) |
| High | XX (XX.X) |
| Visit 3 / Week 4 | |
| n | XX |
| Normal | XX (XX.X) |
| Out of Range | XX (XX.X) |
| Low | XX (XX.X) |
| High | XX (XX.X) |
| Visit 5 / Week 8 | |
| n | XX |
| Normal | XX (XX.X) |
| Out of Range | XX (XX.X) |
| Low | XX (XX.X) |
| High | XX (XX.X) |

N: the number of subjects in the Safety population.

n: the number of subjects within a specific category or number of valid observations. Percentages are based on the corresponding number of valid observations.

<sup>[1]</sup> Number of subjects with at least one non-missing post-baseline assessment of the corresponding parameter.



Similar to table 14.4.2.2.1, the following tables will be constructed:

Table 14.3.4.5.2 Incidence of Blood Chemistry Assessments Outside of Normal Range Table 14.3.4.5.3 Incidence of Morning Urine Assessments Outside of Normal Range



### **Local Skin Reactions Assessment**

MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.6.1 Summary of Local Skin Reactions Assessment

Safety population Page X of X

| sit | Total |
|-------------------------|------------|
| Investigator Assessment | (N = XX) |
| Investigator Assessment | n (%) |
| aseline | |
| n | XX |
| 0 (Absent) | XX (XX.X) |
| 1 (Mild) | XX (XX.X) |
| 2 (Moderate) | XX (XX.X) |
| 3 (Severe) | XX (XX.X) |
| sit 2 / Week 2 | |
| n | XX |
| 0 (Absent) | XX (XX.X) |
| 1 (Mild) | XX (XX.X) |
| 2 (Moderate) | XX (XX.X) |
| 3 (Severe) | XX (XX.XX) |
| sit 3 / Week 4 | |
| n | XX |
| 0 (Absent) | XX (XX.X) |
| 1 (Mild) | XX (XX.X) |
| 2 (Moderate) | XX (XX.X) |
| 3 (Severe) | XX (XX.X) |
| • | |
| • • • | ••• |

N: the number of subjects in the Safety population.

n: the number of subjects within a specific category or the number of valid observations. Percentages are based on the corresponding number of valid observations.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug application.



Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Report the following parameters: Investigator assessment of Erosion/ulceration in lesional area, Vesicles in lesional area, Erythema in perilesional area, Scaling in the perilesional area, Edema in perilesional area, Atrophy in perilesional area, Vesicles in perilesional area, Erosion/ulceration in perilesional area, Subject assessment of Burning or pain after application.

Report the following visits: Baseline, Visit 2 / Week 2, Visit 3 / Week 4, Visit 4 / Week 6, Visit 5 / Week 8, Most severe post-baseline.

### **Programming note:**

For parameter "Subject assessment of Burning or pain after application" report Visit 1/ Day 0 instead of Baseline assessment.



MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.6.2 Local Skin Reactions Assessment Shifts from Baseline

Safety population Page X of X

| | | | Baseline | | |
|---|---|---|---|---|---|
| | 0 (Absent) | 1 (Mild) | 2 (Moderate) | 3 (Severe) | Total |
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| Visit 2 / Week 2 | | | | | |
| 0 (Absent) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 (Mild) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 (Moderate) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 3 (Severe) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Total | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Visit 3 / Week 4 | | | | | |
| ••• | • • • | ••• | ••• | • • • | • • • |
| ••• | | | | | |

N: the number of subjects in the Safety population.

For the most severe post-baseline values percentages are based on the number of subjects with non-missing assessment at baseline and at least one non-missing post-baseline assessment for the corresponding parameter.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Report the following parameters: : Investigator assessment of Erosion/ulceration in lesional area, Vesicles in lesional area, Erythema in perilesional area, Scaling in the perilesional area, Edema in perilesional area, Atrophy in perilesional area, Vesicles in perilesional area, Erosion/ulceration in perilesional area.

Report the following visits: Visit 2 / Week 2, Visit 3 / Week 4, Visit 4 / Week 6, Visit 5 / Week 8, Most severe post-baseline.

n: the number of subjects within a specific category. Percentages are based on the number of non-missing values at baseline and at the corresponding visit.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug application.

Percentages are based on the number of subjects with non-missing assessment at the corresponding time point and at baseline.



MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.6.3 Summary of LSR Sum Score

Safety population Page X of X

| | Total $(N = XX)$ | Change from the baseline |
|------------------|------------------|--------------------------|
| Baseline | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.X | |
| Median | XX.X | |
| Q1, Q3 | XX.X, XX.X | |
| Min, Max | XX, XX | |
| Visit 2 / Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.X | XX.X |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX |
| Visit 3 / Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.X | XX.X |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX |
| ••• | | |

LSR=Local Skin Reactions.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug application.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

N: the number of subjects in the Safety population.

n: the number of valid measurements.





Report the following visits: Visit 2 / Week 2, Visit 3 / Week 4, Visit 4 / Week 6, Visit 5 / Week 8.



Vital signs

MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.7.1 Summary of Vital Signs

Safety population Page X of X

Parameter: XXXXXXXXXXXXX (units)

| | Total $(N = XX)$ | Change from the baseline |
|------------------|------------------|--------------------------|
| Baseline | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.X | |
| Median | XX.X | |
| Q1, Q3 | XX.X, XX.X | |
| Min, Max | XX, XX | |
| Visit 2 / Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.X | XX.X |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX |
| ••• | ••• | |

N: the number of subjects in the Safety population.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

n: the number of valid measurements.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug application.



Report the following parameters: Systolic blood pressure (mm Hg)/ Diastolic blood pressure (mm Hg)/ Pulse rate (beats/minute)/ Oral temperature (C), Tympanic temperature (C).

Report the following visits: Baseline, Visit 2 / Week 2, Visit 3 / Week 4, Visit 4 / Week 6, Visit 5 / Week 8, Highest post-baseline, Lowest post-baseline.



MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.7.2 Incidence of Vital Signs Assessments Outside of Normal Range

Safety population Page X of X

Parameter: XXXXXXXXXXXXX (units)

| | Total<br>(N = XX)<br>n (%) |
|---------------------------------------|----------------------------|
| Any Time After the Start of Treatment | |
| n [1] | XX |
| Out of Range | XX (XX.X) |
| Low | XX (XX.X) |
| High | XX (XX.X) |
| Baseline | |
| n | XX |
| Normal | XX (XX.X) |
| Out of Range | XX (XX.X) |
| Low | XX (XX.X) |
| High | XX (XX.X) |
| Visit 2 / Week 2 | |
| n | XX |
| Normal | XX (XX.X) |
| Out of Range | XX (XX.X) |
| Low | XX (XX.X) |
| High | XX (XX.X) |
| | ••• |

N: the number of subjects in the Safety population.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

n: the number of subjects within a specific category or number of valid observations. Percentages are based on the corresponding number of valid observations.

<sup>[1]</sup> Number of subjects with at least one non-missing post-baseline assessment of the corresponding parameter.



Report the following parameters: Systolic blood pressure (mm Hg)/ Diastolic blood pressure (mm Hg)/ Pulse rate (beats/minute)/ Oral temperature (C), Tympanic temperature (C).

Report the following visits: Any Time After the Start of Treatment, Baseline, Visit 2 / Week 2, Visit 3 / Week 4, Visit 4 / Week 6, Visit 5 / Week 8.



MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.7.3 Incidence of Notably Abnormal Vital Signs Assessments

Safety population Page X of X

Parameter: XXXXXXXXXXXX (units)

| | Total $(N = XX)$ |
|---|---|
| | n (%) |
| Any Time After the Start of Treatment | |
| n [1] | XX |
| Low (90 mmHg or lower and decreased by 20 mmHg or more) | XX (XX.X) |
| High (180 mmHg or greater and increased by 20 mmHg or more) | XX (XX.X) |
| Baseline | |
| n | XX |
| Low (90 mmHg or lower) | XX (XX.X) |
| High (180 mmHg or greater) | XX (XX.X) |
| Visit 2 / Week 2 | |
| n | XX |
| Low (90 mmHg or lower and decreased by 20 mmHg or more) | XX (XX.X) |
| High (180 mmHg or greater and increased by 20 mmHg or more) | XX (XX.X) |
| ••• | ••• |

N: the number of subjects in the Safety population.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Report the following parameters: Systolic blood pressure (mm Hg)/ Diastolic blood pressure (mm Hg)/ Pulse rate (beats/minute). Criteria for notable vital signs measurements are specified in SAP Section 9.5.

Report the following visits: Any Time After the Start of Treatment, Baseline, Visit 2 / Week 2, Visit 3 / Week 4, Visit 4 / Week 6, Visit 5 / Week 8.

n: the number of subjects within a specific category or number of valid observations. Percentages are based on the corresponding number of valid observations.

<sup>[1]</sup> Number of subjects with at least one non-missing post-baseline assessment of the corresponding parameter.



### **Physical Examination**

MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.8 Summary of Physical Parameters

Safety population Page X of X

Parameter: Weight (kg)

| | | Change from the baseline |
|------------------|------------|--------------------------|
| Baseline | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.X | |
| Median | XX.X | |
| Q1, Q3 | XX.X, XX.X | |
| Min, Max | XX, XX | |
| Visit 3 / Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.X | XX.X |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX |
| • • • | ••• | • • • |

N: the number of subjects in the Safety population.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug application.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Report the following parameters: Weight (kg)/ Height (cm)/ BMI (kg/m2). Report the following visits: Baseline, Visit 3 / Week 4, Visit 5 / Week 8.

n: the number of valid measurements.



MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.9 Summary of Physical Examination

Safety population Page X of X

Abbreviated physical examination

| | Total $(N = XX)$ |
|------------------|------------------|
| | n (%) |
| Baseline | |
| n | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | XX (XX.X) |
| Abnormal CS | XX (XX.X) |
| Visit 3 / Week 4 | |
| n | XX |
| Normal | XX (XX.X) |
| Abnormal NCS | xx (xx.x) |
| Abnormal CS | XX (XX.X) |
| ••• | |
| • • • | ••• |

CS=Clinically Significant; NCS=Not clinically significant.

N: the number of subjects in the Safety population.

n: the number of subjects within a specific category or number of valid observations. Percentages are based on the corresponding number of valid observations.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Repeat for Complete dermatological examination.

Report the following visits: Baseline, Visit 3 / Week 4, Visit 5 / Week 8, Follow-up.





**ECG** 

MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.10.1 Summary of Electrocardiogram

Safety population Page X of X

Parameter: XXXXXXXXXXXXXX (units)

| | Total Change $(N = XX)$ the bas | |
|------------------|---------------------------------|------|
| Baseline | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.X | |
| Median | XX.X | |
| Q1, Q3 | XX.X, XX.X | |
| Min, Max | XX, XX | |
| Visit 3 / Week 4 | | |
| n | XX XX | X |
| Mean | XX.X XX. | . X |
| SD | XX.X XX. | . X |
| Median | XX.X XX. | . X |
| Q1, Q3 | XX.X, XX.X XX.X, | XX.X |
| Min, Max | XX, XX XX, | XX |
| Visit 5 / Week 8 | | |
| n | XX XX | X |
| Mean | XX.X XX. | . X |
| SD | XX.X XX. | |
| Median | XX.X XX. | . X |
| Q1, Q3 | XX.X, XX.X XX.X, | |
| Min, Max | XX, XX XX, | |
| ••• | ••• | |

QTC-F=QT interval corrected according to Fridericia's formula; QTC-B=QT interval corrected according to Bazett's formula. N: the number of subjects in the Safety population.



n: the number of valid measurements.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug application.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Report the following parameters: Heart rate (beats/min)/ RR interval (msec)/ PR interval (msec)/ QRS duration (msec), QT interval (msec), QTC-F interval (msec), QTC-B interval (msec).

Report the following visits: Baseline, Visit 3 / Week 4, Visit 5 / Week 8, Highest post-baseline, Lowest post-baseline.



MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.10.2 Incidence of Abnormal ECG Assessments

Safety population Page X of X

Parameter: General Assessment

| | Total<br>(N = XX)<br>n (%) | |
|---|---|---|
| Any Time After the Start of Treatment | | |
| n [1] | | XX |
| Abnormal | XX | (XX.X) |
| Abnormal CS | | (XX.X) |
| Baseline | | |
| n | | XX |
| Normal | XX | (XX.X) |
| Abnormal NCS | XX | (XX.X) |
| Abnormal CS | XX | (XX.X) |
| Visit 3 / Week 4 | | |
| n | | XX |
| Normal | XX | (XX.X) |
| Abnormal NCS | XX | (XX.X) |
| Abnormal CS | XX | (XX.X) |
| Visit 5 / Week 8 | | |
| n | | XX |
| Normal | XX | (XX.X) |
| Abnormal NCS | XX | (XX.X) |
| Abnormal CS | | (XX.X) |
| | | ••• |

N: the number of subjects in the Safety population. n: the number of subjects within a specific category or number of valid observations. Percentages are based on the corresponding number of valid observations.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

<sup>[1]</sup> Number of subjects with at least one non-missing post-baseline assessment of the corresponding parameter.



### **Programming note:**

Report the following visits: Any Time After the Start of Treatment, Baseline, Visit 3 / Week 4, Visit 5 / Week 8.



MC2 Therapeutics MC2-01-C6

#### Table 14.3.4.10.3 Incidence of Notably Abnormal ECG Assessments

Safety population Page X of X

Parameter: XXXXXXXXXXXXX (units)

| | Total |
|------------------------------------------|-------------------|
| | (N = XX)<br>n (%) |
| | 11 (%) |
| Any Time After the Start of Treatment | |
| n [1] | XX |
| QTc interval > 450 | XX (XX.X) |
| QTc interval > 480 | XX (XX.X) |
| QTc interval > 500 | XX (XX.X) |
| QTc interval increases from baseline >30 | XX (XX.X) |
| QTc interval increases from baseline >60 | XX (XX.X) |
| Baseline | |
| n | XX |
| QTc interval > 450 | XX (XX.X) |
| QTc interval > 480 | XX (XX.X) |
| QTc interval > 500 | XX (XX.X) |
| Visit 3 / Week 4 | |
| n | XX |
| QTc interval > 450 | XX (XX.X) |
| QTc interval > 480 | XX (XX.X) |
| QTc interval > 500 | XX (XX.X) |
| QTc interval increases from baseline >30 | XX (XX.X) |
| QTc interval increases from baseline >60 | XX (XX.X) |
| ••• | |
| ••• | ••• |

N: the number of subjects in the Safety population.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

ma+a1

n: the number of subjects within a specific category or number of valid observations. Percentages are based on the corresponding number of valid observations.

<sup>[1]</sup> Number of subjects with at least one non-missing post-baseline assessment of the corresponding parameter.



### **Programming note:**

Report the following parameters: QTC-F interval (msec), QTC-B interval (msec).

Report the following visits: Any Time After the Start of Treatment, Baseline, Visit 3 / Week 4, Visit 5 / Week 8.





### Physician Global Assessment of Psoriasis Severity

MC2 Therapeutics MC2-01-C6

#### Table 14.4.1.1 Summary of PGA

Safety population Page X of X

| /isit | | Change from baseline |
|------------------|------------|----------------------|
| Baseline | | |
| n | XX | |
| Mean | XX.X | |
| SD | XX.X | |
| Median | XX.X | |
| Q1, Q3 | XX.X, XX.X | |
| Min, Max | XX, XX | |
| 7isit 2 / Week 2 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.X | XX.X |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX |
| /isit 3 / Week 4 | | |
| n | XX | XX |
| Mean | XX.X | XX.X |
| SD | XX.X | XX.X |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| Min, Max | XX, XX | XX, XX |
| • | , | , |
| ••• | | |

PGA=Physician global assessment.

N: the number of subjects in the Safety population.

n: the number of valid observations.



Baseline is the last non-missing assessment prior to the first dose of the study drug.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Report the following visits: Baseline, Visit 2 / Week 2, Visit 3 / Week 4, Visit 4 / Week 6, Visit 5 / Week 8.



MC2 Therapeutics MC2-01-C6

#### Table 14.4.1.2 Summary of Treatment Success

Safety population Page X of X

| | | Total<br>(N = XX) |
|-------------------|-------------------------|-------------------------|
| | | , |
| Treatment success | | |
| Overall | n' (%) [1]<br>n (%) [2] | XX (XX.X)<br>XX (XX.X) |
| | 95% CI | XX.X, XX.X |
| Visit 2 / Week 2 | n' (%) [1] | XX (XX.X) |
| | n (%) [2]<br>95% CI | XX (XX.X)<br>XX.X, XX.X |
| Visit 3 / Week 4 | n' (%) [1] | XX (XX.X) |
| | n (%) [2]<br>95% CI | XX (XX.X)<br>XX.X, XX.X |
| | 93% C1 | ΛΛ.Α, ΛΛ.Λ |
| ••• | ••• | ••• |

PGA=Physician global assessment.

N: the number of subjects in the Safety population. n: the number of subjects within a specific category. n': the number of valid observations.

Treatment success is defined as at least 2-point decrease from Baseline in the PGA on the trunk, limbs, and scalp.

Baseline is the last non-missing assessment prior to the first dose of the study drug. Only subjects having at least moderate severity at baseline will be included into the summary.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Report the following visits: Overall, Visit 2 / Week 2, Visit 3 / Week 4, Visit 4 / Week 6, Visit 5 / Week 8.

<sup>[1]</sup> Subjects having any post-baseline values (for 'Overall' category) or values at the corresponding visit. Percentage is calculated as (100 x n/N).

<sup>[2]</sup> Percentages are based on the corresponding number of valid observations.

Confidence interval is calculated using Clopper-Pearson method.



MC2 Therapeutics MC2-01-C6

#### Table 14.4.1.3 PGA Shifts from Baseline

Safety population Page X of X

| | | Baseline | | | | | |
|---|---|---|---|---|---|---|---|
| | | 0 - Clear | 1 - Almost Clear | 2 - Mild | 3 - Moderate | 4 - Severe | Total |
| Visit 2 / Week 2 | | | | | | | |
| 0 - Clear | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| 1 - Almost Clear | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 2 - Mild | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| 3 - Moderate | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| 4 - Severe | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| Total | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |
| Visit 3 / Week 4 | | | | | | | |
| 0 - Clear | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| 1 - Almost Clear | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| 2 - Mild | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| 3 - Moderate | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| 4 - Severe | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X |
| Total | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (100) |

PGA=Physician global assessment.

The baseline value for a variable is defined as the last non-missing value collected before the first study drug application. Percentages are based on the number of subjects with non-missing assessment at the corresponding time point and at baseline.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings



### **Body Surface Area Involvement Assessment**

MC2 Therapeutics MC2-01-C6

#### Table 14.4.2.1 Summary of Body Surface Area Involvement

Safety population Page X of X

Parameter: XXXXXXXXXXXXXXXX (%)

| | | Change from the baseline |
|------------------|--------------|--------------------------|
| Baseline | | |
| n | XX | |
| Mean | XX.XX | |
| SD | XX.XX | |
| Median | XX.XX | |
| Q1, Q3 | XX.XX, XX.XX | |
| Min, Max | XX.X, XX.X | |
| Visit 3 / Week 4 | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |
| Visit 5 / Week 8 | | |
| n | XX | XX |
| Mean | XX.XX | XX.XX |
| SD | XX.XX | XX.XX |
| Median | XX.XX | XX.XX |
| Q1, Q3 | XX.XX, XX.XX | XX.XX, XX.XX |
| Min, Max | XX.X, XX.X | XX.X, XX.X |

BSA=Body Surface Area.

N: the number of subjects in the Safety population.

n: the number of valid measurements.



The baseline value for a variable is defined as the last non-missing value collected before the first study drug application.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

### **Programming note:**

Report the following parameters: Scalp BSA psoriatic involvement (%), Neck, Trunk and/or Limbs BSA psoriatic involvement (%), Total psoriatic involvement (%).

Report the following visits: Baseline, Visit 3 / Week 4, Visit 5 / Week 8.



### **Psoriasis Treatment Convenience Scale**

MC2 Therapeutics MC2-01-C6

#### Table 14.4.3.1 Summary of Psoriasis Treatment Convenience Scale

Safety population Page X of X

Parameter: XXXXXXXXXXXXXXXXX

| | Total |
|------------------|------------|
| | (N = XX) |
| Visit 2 / Week 2 | |
| n | XX |
| Mean | XX.X |
| SD | XX.X |
| Median | XX.X |
| Q1, Q3 | xx.x, xx.x |
| Min, Max | XX, XX |
| Visit 3 / Week 4 | |
| n | XX |
| Mean | xx.x |
| SD | XX.X |
| Median | xx.x |
| Q1, Q3 | XX.X, XX.X |
| Min, Max | XX, XX |
| Titi, Tak | , |
| ••• | |
| ••• | ••• |

PTCS=Psoriasis Treatment Convenience Scale.

N: the number of subjects in the Safety population.

Each question is rated on a 1-10 scale from least to most favorable response. PTCS total score is the sum of the scores on questions 1 to 5. If more than two questions are not answered, the PTCS total score is missing. If one or two questions remain unanswered, the missing scores are replaced by the average of the answered scores for the summation.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

n: the number of valid measurements.



### **Programming note:**

Report the following parameters: PTCS Total Score, Q1. How easy was the treatment to apply to the skin?, Q2. How greasy was the treatment when applying it to the skin?, Q3. How moisturized did your skin feel after applying the treatment?, Q4. How greasy did your skin feel after applying the treatment?, Q5. How much did treating your skin disrupt your daily routine?, Q6. Overall, how satisfied were you with the medical treatment?.

Report the following visits: Visit 2 / Week 2, Visit 3 / Week 4, Visit 5 / Week 8.



**Figures Shells** 

MC2 Therapeutics MC2-01-C6

Figure 16.2.5.4 Individual BDP Plasma Concentration-time Profiles on Linear and Semi-logarithmic Scales Week 4

PK population
Subject=XXXX







BDP=Betamethasone dipropionate; BLQ=Below Limit of Quantification; LLOQ=Lower Limit of Quantification.
BLQ concentrations were substituted with LLOQ for the calculation for graphic presentation. LLOQ for BDP is XX.X pq/mL.

Path to the program code, date and time of output/ Datasets used/ Referenced Data Listings

Similar to figure 16.2.5.4, the following figures will be constructed (with modification of underlined fragments):

Figure 16.2.5.5 Individual Calcipotriol (CAL) Plasma Concentration-time Profiles on Linear and Semi-logarithmic Scales Week 4
Figure 16.2.5.6 individual MC1080 Plasma Concentration-time Profiles on Linear and Semi-logarithmic Scales Week 4
Figure 16.2.5.7 individual Betamethasone 17-propionate, Plasma Concentration-time Profiles on Linear and Semi-logarithmic Scales Week 4



**Listings Shells** 

MC2 Therapeutics MC2-01-C6

#### Listing 16.2.1.1 Analysis Populations

All Enrolled subjects Page X of X

| Country/Site ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | All<br>Enrolled<br>subjects | Date of Informed<br>Consent/Assent | Allocated<br>to<br>treatment | Safety<br>Population | HPA<br>Population | Reason for<br>Exclusion<br>from HPA<br>population | PK<br>Population | Reason for<br>Exclusion<br>from PK<br>population |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | Yes | YYYY-MM-DD/ XX/<br>YYYY-MM-DD/ XX | No | No | No | XXXXXXXXX | No | XXXXXXXXX |
| XXX/XX/XXXXX | 15/M/W/HL | Yes | YYYY-MM-DD/ XX/<br>YYYY-MM-DD/ XX | Yes | Yes | Yes | | No | XXXXXXXXX |
| XXX/XX/XXXXX | 16/F/A/NHL | Yes | YYYY-MM-DD/ XX/<br>YYYY-MM-DD/ XX | Yes | Yes | Yes | | Yes | |
| | | | YYYY-MM-DD/ XX | | | | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. HPA=Hypothalamic-pituitary-adrenal; PK=Pharmacokinetics.

Path to the program code, date and time of output/ Datasets used



MC2 Therapeutics MC2-01-C6

Listing 16.2.1.2 Subject Visits

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Visit | Date / Study day | Main reason for unscheduled visit |
|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXXX | YYYY-MM-DD/ XX | |
| XXX/XX/XXXXX | 15/M/W/HL | XXXXXX | YYYY-MM-DD/ XX | |
| XXX/XX/XXXXX | 16/F/A/NHL | XXXXXX | YYYY-MM-DD/ XX | XXXXXXXXXX XXXXXXXXXX |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

Path to the program code, date and time of output/ Datasets used



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.1.3 Study Completion

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject ID | Age(Years)/<br>Sex/Race/ | Date of Study Completion or Discontinuation/ Study Day | End of Study<br>Status | Reason for Study Discontinuation |
|---|---|---|---|---|
| | Ethnicity | | | |
| XXX/XX/XXXXX | 14/F/A/NHL | YYYY-MM-DD/ XX | Discontinued | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX/XX/XXXXX | 15/M/W/HL | YYYY-MM-DD/ XX | Discontinued | Other: XXXXXXXXXXXXXXXXXXXXX |
| XXX/XX/XXXXX | 16/F/A/NHL | YYYY-MM-DD/ XX | Completed | |
| XXX/XX/XXXXX | 16/M/A/NHL | YYYY-MM-DD/ XX | Screening failure | Inconsistency with inclusion / exclusion criteria: XXXXX |

. . .

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

Path to the program code, date and time of output/ Datasets used


MC2 Therapeutics MC2-01-C6

### Listing 16.2.1.4 Study Treatment Completion

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Date of Study Treatment<br>Completion or<br>Discontinuation/ Study Day | Was the IP<br>discontinued before<br>Week 8 visit? | Reason for Study Treatment Discontinuation |
|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | YYYY-MM-DD/ XX | Yes | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| XXX/XX/XXXXX | 15/M/W/HL | YYYY-MM-DD/ XX | Yes | Other: XXXXXXXXXXXXXXXXXXXX |
| XXX/XX/XXXXX | 16/F/A/NHL | YYYY-MM-DD/ XX | No | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.



MC2 Therapeutics MC2-01-C6

### Listing 16.2.2.1 Violation of Inclusion/Exclusion Criteria

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Category | Criterion number/Criterion | Result |
|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | Inclusion criteria | XX/XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | No |
| | | Exclusion criteria | XX/XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes |
| | | Exclusion criteria | XX/XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Yes |
| • • • | | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.2.2 Protocol Deviations

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject<br>ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Date of<br>Deviation<br>Revealed | Visit | Deviation Category/<br>Subcategory | Issue | Description of deviation | Assessment |
|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | YYYY-MM-DD | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Major |
| XXX/XX/XXXXX | 15/M/W/HL | YYYY-MM-DD | XXXXX | XXXXXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Minor |
| XXX/XX/XXXXX | 16/F/A/NHL | YYYY-MM-DD | XXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Minor |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.4.1 Demographics and Other Baseline Characteristics

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject | Age(Years)/<br>Sex/Race/ | Year of<br>Birth | Fitzpatrick Skin<br>Type | Date of<br>Diagnosis | Duration of<br>Disease (months) | Previous Treatments |
|---|---|---|---|---|---|---|
| ID | Ethnicity | | | | | |
| XXX/XX/XXXXX | 14/F/A/NHL | YYYY | XXXXXXXXXXXX | YYYY-MM | XX.X | Systemic: Biologics and systemic/ TNF-a inhibitors/ Topical: vitamin D analogs |
| XXX/XX/XXXXX | 15/M/W/HL | YYYY | XXXXXXXXXXXXX | YYYY-MM | XX.X | |
| XXX/XX/XXXXX | 16/F/A/NHL | YYYY | XXXXXXXXXXXXX | YYYY-MM | XX.X | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.4.2 Baseline Variables

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter | (Unit) | Visit | Result |
|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXXXXXX | (XXXXXX) | Scr V1 | XX.X |
| | | | | Scr V2 | XX.X |
| | | | | V1 Day0 | XX.X |
| | | | | Baseline | XX.X |
| | | XXXXXXXXX | (XXXXXX) | Scr V1 | XX.X |
| | | | | Scr V2 | XX.X |
| | | | | | ••• |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.4.3 Medical History

All Enrolled subjects
Page X of X

| Country/Site ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | System Organ Class/<br>Preferred Term/<br>Lowest Level Term/<br>Condition/Diagnosis | Prior/Concurrent | Start Date/<br>Study Day | End Date /<br>Study Day | Ongoing at the End<br>of Clinical Trial |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | PR | YYYY-MM-DD/<br>XX | YYYY-MM-DD/ XX | Resolved |

 ${\tt Country: CZE=Czech \ Republic, \ HUN=Hungary, \ DEU=Germany; \ Sex: \ F=Female, \ M=Male;}$ 

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

PR=Prior, C=Concomitant.

Terms are coded by MedDRA version XX.X.

Path to the program code, date and time of output/ Datasets used

### **Programming note:**

Sort by ascending start date within subject.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.4.4 Prior/Concomitant Therapy

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject<br>ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | 3rd Lvl, Pharmacological Subgroup/<br>4th Lvl, Chemical Subgroup/<br>5th Lvl, Chemical Substance/<br>Medication | Prior/<br>Concomitant | Start Date/<br>Study Day/<br>Stop Date/<br>Study Day | Dose (Units)/<br>Frequency/<br>Route | Formulation/<br>Location | Indication |
|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | PR | YYYY-MM-DD/<br>XX/<br>YYYY-MM-DD/<br>XX | XXXXX (XXXXX) /<br>XXXXX/<br>XXXXX | XXXXX/<br>XXXXX | XXXXXXXXXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | С | YYYY-MM-DD/<br>XX/<br>Ongoing | XXXXX (XXXXX)/<br>XXXXX/<br>XXXXX | XXXXX/<br>XXXXX | xxxxxxxxxx |

...

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

PR=Prior, C=Concomitant, PT=Post-Treatment.

Drug and non-drug therapy records are coded using WHODD version XX.X.

Path to the program code, date and time of output/ Datasets used

### **Programming note:**

Sort by ascending start date within subject.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.4.5 Prior/Concomitant Procedures

All Enrolled subjects
Page X of X

| Country/Site ID/ | Age(Years)/ | System Organ Class/ | Start date, Time/ | Location | Indication |
|---|---|---|---|---|---|
| ubject ID | Sex/Race/ | Preferred Term/ | Study day/ | | |
| | Ethnicity | Lowest Level Term/ | Stop date, Time/ | | |
| | | Therapy/Procedure | Study day | | |
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD HH:MM/ XX/ | XXXXXXXXXXXXX | XXXXXXXXXX |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD HH:MM/ XX | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | |
| | | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. Procedures are coded using MedDRA version XX.X.

Path to the program code, date and time of output/ Datasets used

### **Programming note:**

Sort by ascending start date within subject.



MC2 Therapeutics MC2-01-C6

### Listing 16.2.5.1 Exposure

Safety population Page X of X

| Country/Site<br>ID/ Subject<br>ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Study Period | Date of First<br>Application/<br>Study Day | Date of Last<br>Application/<br>Study Day | Total Duration of Exposure (days) | Extent of<br>Exposure<br>(days) | Number<br>of<br>Missed<br>Doses | Total Dose (g)/<br>Average Weekly<br>Dose (g) | Compliance (%) |
|---|---|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | Overall | YYYY-MM-DD/ 1 | YYYY-MM-DD/ XX | XX | XX | XX | XX.X/ XX.X | XX.X |
| | | Up to Week 2 | YYYY-MM-DD/ 1 | YYYY-MM-DD/ XX | XX | XX | XX | XX.X/ XX.X | XX.X |
| | | Up to Week 4 | YYYY-MM-DD/ 1 | YYYY-MM-DD/ XX | XX | XX | XX | XX.X/ XX.X | XX.X |
| | | From Week 4<br>to Week 8 | YYYY-MM-DD/<br>XX | YYYY-MM-DD/ XX | XX | XX | XX | XX.X/ XX.X | XX.X |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. Lost and unused tubes were not accounted for in the calculation of total dose.



MC2 Therapeutics

### Listing 16.2.5.2 Study Drug Compliance

Safety population Page X of X

| Country/Site ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Visit | Was the subject<br>diary completed by<br>the patient<br>(Reason, if Not<br>Completed)? | Did the subject apply<br>the study drug once<br>daily to the scalp,<br>trunk and/or limbs<br>since the last visit? | Is the PGA "clear" and was the subject recommended to stop the treatment with study drug at the visit? | Was the treatment with study drug restarted by the subject after interruption at the last visit?/ Restart Date |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | V2/Week2 | | XXX | | |
| | | V3/Week4 | XXX | XXX | XXX | |
| | | V5/Week8 | XXX | XXX | | XXX/ YYYY-MM-DD |
| | | • • • | • • • | ••• | | ••• |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.5.3 Missed Doses

Safety population Page X of X

| Country/Site ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Date/ Study Day | Reason Not Administered |
|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | YYYY-MM-DD/ XX | Approved Discontinuation |
| | | YYYY-MM-DD/ XX | Missed |
| | | YYYY-MM-DD/ XX | Missed |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.5.4 Study Drug Accountability

Allocated to treatment Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Visit<br>Dispensed | Kit Number | Date Dispensed/ Study Day/<br>Date Returned/ Study Day | Tube Assessment | Returned<br>Amount | Used Between |
|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | V1 (Day 0) | XXXXXXXX | YYYY-MM-DD/ XX/<br>YYYY-MM-DD/ XX/ | SEAL BROKEN | XX.X g | xxxxxxxxxxx/<br>xxxxxxxxxxxx |
| | | | XXXXXXXX | YYYY-MM-DD/ XX/<br>YYYY-MM-DD/ XX/ | SEALED | | |
| | | | xxxxxxxx | YYYY-MM-DD/ XX/<br>YYYY-MM-DD/ XX/ | SEAL BROKEN | XX.X g | XXXXXXXXXXXX/<br>XXXXXXXXXXXX |

. . .

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.7.1 Adverse Events

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject<br>ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | AE<br>No/<br>TEAE<br>[1]/<br>SAE<br>[2] | System Organ Class/<br>Preferred Term/<br>Lowest Level Term/<br>Reported Term | Start Date, Time/<br>Study Day/<br>End Date, Time/<br>Study Day | Severity/ Relationship to IP/ Action taken with IP/ Outcome | Concomitant therapy?/ Concomitant non-drug therapy?/ Concomitant procedures?/ Did subject withdraw due to this AE?/ Is AE related to Cosyntropin?/ Is AE related to a study procedure (specify)? Location of AE to Treatment Area |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XX/<br>XXX/<br>XXX<br>(X,X) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD HH:MM/<br>XXX/<br>YYYY-MM-DD HH:MM/<br>XXX | XXXXXXXXX/<br>XXXXXXXXX/<br>XXXXXXXXXX/<br>XXXXXX | XXX/ XXX/ XXX/<br>XXX/ XXX (XXXXXXXX XXXXXXXXX)/<br>XXXXXXXXXXXXXX |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

AE = Adverse Event, SAE = Serious Adverse Event, TEAE = Treatment-Emergent Adverse Event; IP=Investigational Product.

AEs are coded using MedDRA version XX.X.

<sup>[1]</sup> TEAE is any reported adverse event that starts after initiation of the study therapy.

<sup>[2]</sup> Seriousness criteria: 1 = <<Death>>, 2 = <<Life-threatening>>, 3 = <<Requires in-patient hospitalization or prolongation of existing hospitalization>>, 4 = << Results in persistent or significant disability/incapacity>>, 5 = << Congenital anomaly/birth defect>>, 6 = << Other serious or important medical event>>.



MC2 Therapeutics MC2-01-C6

### Listing 16.2.7.2 Serious Adverse Events

All Enrolled subjects Page X of X

| Country/Site<br>ID/ Subject<br>ID | Age(Years)<br>/<br>Sex/Race/<br>Ethnicity | AE No/<br>TEAE<br>[1]/<br>SAE<br>[2] | System Organ Class/<br>Preferred Term/<br>Lowest Level Term/<br>Reported Term | Start Date, Time/<br>Study Day/<br>End Date, Time/<br>Study Day | Severity/ Relationship to IP/ Action taken with IP/ Outcome | Concomitant therapy?/ Concomitant non-drug therapy?/ Concomitant procedures?/ Did subject withdraw due to this AE?/ Is AE related to Cosyntropin?/ Is AE related to a study procedure (specify)?/ Location of AE to Treatment Area |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XX/<br>XXX/<br>XXX<br>(X,X) | ************************************** | YYYY-MM-DD HH:MM/<br>XXX/<br>YYYY-MM-DD HH:MM/<br>XXX | xxxxxxxxx/<br>xxxxxxxxxx/<br>xxxxxxxxxx/<br>xxxxxx | XXX/ XXX/ XXX/<br>XXX/ XXX/ XXX (XXXXXXXX XXXXXXXXX)/<br>XXXXXXXXXXXXXX |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

AE = Adverse Event, SAE = Serious Adverse Event, TEAE = Treatment-Emergent Adverse Event; IP=Investigational Product.

AEs are coded using MedDRA version XX.X.

<sup>[1]</sup> TEAE is any reported adverse event that starts after initiation of the study therapy.

<sup>[2]</sup> Seriousness criteria: 1 = <<Death>>, 2 = <<Life-threatening>>, 3 = << Requires in-patient hospitalization or prolongation of existing hospitalization>>, 4 = << Results in persistent or significant disability/incapacity>>, 5 = << Congenital anomaly/birth defect>>, 6 = << Other serious or important medical



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.7.3 Listing of Adverse Events Leading Discontinuation of Study Drug

Safety population Page X of X

| Country/Site<br>ID/ Subject<br>ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | AE<br>No/<br>TEAE<br>[1]/<br>SAE<br>[2] | System Organ Class/<br>Preferred Term/<br>Lowest Level Term/<br>Reported Term | Start Date, Time/<br>Study Day/<br>End Date, Time/<br>Study Day | Severity/ Relationship to IP/ Action taken with IP/ Outcome | Concomitant therapy?/ Concomitant non-drug therapy?/ Concomitant procedures?/ Did subject withdraw due to this AE?/ Is AE related to Cosyntropin?/ Is AE related to a study procedure (specify)?/ Location of AE to Treatment Area |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XX/<br>XXX/<br>XXX<br>(X,X) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD HH:MM/<br>XXX/<br>YYYY-MM-DD HH:MM/<br>XXX | xxxxxxxxx/<br>xxxxxxxxxx/<br>xxxxxxxxxx/<br>xxxxxx | XXX/ XXX/ XXX/<br>XXX/ XXX/ XXX (XXXXXXXX XXXXXXXXX)/<br>XXXXXXXXXXXXXX |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

AE = Adverse Event, SAE = Serious Adverse Event, TEAE = Treatment-Emergent Adverse Event; IP=Investigational Product.

AEs are coded using MedDRA version XX.X.

<sup>[1]</sup> TEAE is any reported adverse event that starts after initiation of the study therapy.

<sup>[2]</sup> Seriousness criteria: 1 = <<Death>>, 2 = <<Life-threatening>>, 3 = <<Requires in-patient hospitalization or prolongation of existing hospitalization>>, 4 = << Results in persistent or significant disability/incapacity>>, 5 = << Congenital anomaly/birth defect>>, 6 = << Other serious or important medical event>>.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.7.4 Listing of Adverse Events Leading to Withdrawal

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject<br>ID | Age (Years) /<br>Sex/Race/<br>Ethnicity | AE<br>No/<br>TEAE<br>[1]/<br>SAE<br>[2] | System Organ Class/<br>Preferred Term/<br>Lowest Level Term/<br>Reported Term | Start Date, Time/<br>Study Day/<br>End Date, Time/<br>Study Day | Severity/ Relationship to IP/ Action taken with IP/ Outcome | Concomitant therapy?/ Concomitant non-drug therapy?/ Concomitant procedures?/ Did subject withdraw due to this AE?/ Is AE related to Cosyntropin?/ Is AE related to a study procedure (specify)?/ Location of AE to Treatment Area |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XX/<br>XXX/<br>XXX<br>(X,X) | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | YYYY-MM-DD HH:MM/<br>XXX/<br>YYYY-MM-DD HH:MM/<br>XXX | XXXXXXXXX/<br>XXXXXXXXX/<br>XXXXXXXXX/<br>XXXXXXX | XXX/ XXX/ XXX/ Yes/ XXX (XXXXXXXX XXXXXXXXX)/ XXXXXXXXXXXXXX |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

AE = Adverse Event, SAE = Serious Adverse Event, TEAE = Treatment-Emergent Adverse Event; IP=Investigational Product.

AEs are coded using MedDRA version XX.X.

<sup>[1]</sup> TEAE is any reported adverse event that starts after initiation of the study therapy.

<sup>[2]</sup> Seriousness criteria: 1 = <<Death>>, 2 = <<Life-threatening>>, 3 = <<Requires in-patient hospitalization or prolongation of existing hospitalization>>, 4 = << Results in persistent or significant disability/incapacity>>, 5 = << Congenital anomaly/birth defect>>, 6 = << Other serious or important medical



MC2 Therapeutics MC2-01-C6

### Listing 16.2.8.1 Hematology in SI Units

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter<br>(Units) | Visit | Date/ Study Day | Result | Reference<br>Range | Change from<br>Baseline | Reason if Not<br>Done/ Comment |
|---|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXX (XXX) | Scr V2 | YYYY-MM-DD/ XX | XX.X @L | XX.X-XX.X | | |
| | | | V3/Week4 | YYYY-MM-DD/ XX | XX.X L | XX.X-XX.X | XX.X | |
| | | | V5/Week8 | | Not Done | XX.X-XX.X | | XXXXXXX XXXXXXX |
| | | | • • • | | | | | |
| | | XXXXX (XXX) | Scr V2 | YYYY-MM-DD/ XX | XX.X @ | XX.X-XX.X | | |
| | | | V3/Week4 | YYYY-MM-DD/ XX | XX.X H | XX.X-XX.X | XX.X | XXXXXXXXXXXXXX |
| | | | V5/Week | YYYY-MM-DD/ XX | XX.X H | XX.X-XX.X | XX.X | |
| • • • | | | • • • | | | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

L = below lower reference limit. H = above upper reference limit.

<sup>@</sup> indicates baseline assessment.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

### Listing 16.2.8.2 Serum Biochemistry in SI Units

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter<br>(Units) | Visit | Date/ Study Day | Result | Reference Range | Change from<br>Baseline | Reason if Not<br>Done/ Comment |
|---|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXX (XXX) | Scr V2<br>V3/Week4<br>V5/Week8 | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | XX.X @L<br>XX.X L<br>Not Done | XX.X-XX.X<br>XX.X-XX.X<br>XX.X-XX.X | XX.X | XXXXXXX XXXXXXX |
| | | XXXXX (XXX) | Scr V2<br>V3/Week4<br>V5/Week | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | XX.X @H<br>XX.X H<br>XX.X H | XX.X-XX.X<br>XX.X-XX.X<br>XX.X-XX.X | xx.x<br>xx.x | xxxxxxxxxx |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

L = below lower reference limit. H = above upper reference limit.

<sup>@</sup> indicates baseline assessment.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.8.3 Morning Urine Assessment in SI Units

All Enrolled subjects
Page X of X

| Country/Site ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter<br>(Units) | Visit | Date/ Study Day | Result | Reference Range | Change from<br>Baseline | Reason if Not<br>Done/ Comment |
|---|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXX (XXX) | Scr V2 | YYYY-MM-DD/ XX | XX.X @L | XX.X-XX.X | | |
| | | | V3/Week4 | YYYY-MM-DD/ XX | XX.X L | XX.X-XX.X | XX.X | |
| | | | V4/Week6 | | Not | XX.X-XX.X | | XXXXXXX XXXXXXX |
| | | | | | Done | | | |
| | | | • • • | | | | | |
| | | XXXXX (XXX) | Scr V2 | YYYY-MM-DD/ XX | XX.X @ | XX.X-XX.X | | |
| | | | V3/Week4 | YYYY-MM-DD/ XX | XX.X L | XX.X-XX.X | XX.X | |
| | | | V4/Week6 | YYYY-MM-DD/ XX | XX.X L | XX.X-XX.X | XX.X | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

L = below lower reference limit. H = above upper reference limit.

<sup>@</sup> indicates baseline assessment.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.8.4 24-hour Urine Assessment

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter<br>(Units) | Visit | Date/ Study Day | Result | Reference Range | Reason if Not<br>Done/ Comment |
|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXX (XXX) | XXXXXXXX | YYYY-MM-DD/ XX | XX.X L | XX.X-XX.X | |
| | | | XXXXXXX | YYYY-MM-DD/ XX | XX.X L | XX.X-XX.X | |
| | | | XXXXXXXX | | Not Done | XX.X-XX.X | XXXXXXX XXXXXXX |
| | | | • • • | | | | |
| | | XXXXX (XXX) | XXXXXXXX | YYYY-MM-DD/ XX | XX.X | XX.X-XX.X | |
| | | | XXXXXXX | YYYY-MM-DD/ XX | XX.X H | XX.X-XX.X | |
| | | | XXXXXXXX | YYYY-MM-DD/ XX | XX.X | XX.X-XX.X | |
| • • • | | | | | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

 ${\tt L}$  = below lower reference limit. H = above upper reference limit.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.8.5 Serum Pregnancy Test

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter<br>(Units) | Visit | Date of Sample/ Study Day | Result | Reasons if Not Done |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXX (XXX) | Scr V2<br>V3/Week4 | YYYY-MM-DD/ XX | XX.X<br>Not Done | XXXXXX XXXXXXXX XXXX |
| | | | V5/Week8 | YYYY-MM-DD/ XX | XX.X | |
| ••• | | | • • • | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. ^ indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.8.6 Urine Pregnancy Test

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Visit | Result | Reasons if Not Done |
|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | Scr V2<br>V3/Week4<br>V5/Week8 | Negative<br>Not Done<br>Negative | XXXXXX XXXXXXXX XXXX |
| ••• | | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. ^ indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.8.7 ACTH Challenge Test

All Enrolled subjects
Page X of X

| Country/Site | Age(Years)/ | Visit | Date, Time of | Parameter (Units) | HPA Axis | Result | Reason if |
|---|---|---|---|---|---|---|---|
| ID/ Subject ID | Sex/Race/ | | assessment/ | | Suppression | | Not Done |
| | Ethnicity | | Study Day | | Noted | | |
| XXX/XX/XXXXX 1 | 14/F/A/NHL | Scr V2 | YYYY-MM-DD | Serum cortisol pre-stimulation | | XX.X | |
| | | | HH:MM/ XX | (nmol/L) | | | |
| | | | YYYY-MM-DD | Serum cortisol post-stimulation | No | XX.X | |
| | | | HH:MM/ XX | (nmol/L) | | | |
| | | V3/Week 4 | YYYY-MM-DD | Serum cortisol pre-stimulation | | XX.X | |
| | | | HH:MM/ XX | (nmol/L) | | | |
| | | | YYYY-MM-DD | Serum cortisol post-stimulation | No | XX.X | |
| | | | HH:MM/ XX | (nmol/L) | | | |
| | | V5/Week 8 | YYYY-MM-DD | Serum cortisol pre-stimulation | | XX.X | |
| | | | HH:MM/ XX | (nmol/L) | | | |
| | | | YYYY-MM-DD | Serum cortisol post-stimulation | No | XX.X | |
| | | | HH:MM/ XX | (nmol/L) | | | |
| | | FU | YYYY-MM-DD | Serum cortisol pre-stimulation | | XX.X | |
| | | | HH:MM/ XX | (nmol/L) | | | |
| | | | YYYY-MM-DD | Serum cortisol post-stimulation | No | XX.X | |
| | | | HH:MM/ XX | (nmol/L) | | | |
| | | | - | • | | | |
| | | | | • • • | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. ^ indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.8.8 Clinically Significant Laboratory Abnormalities

Safety population Page X of X

| Country/Site ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Panel | Visit | Date/ Study Day | Comments |
|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | Hematology<br>XXXXXXXX | V3/Week4<br>V5/Week 8 | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | XXXXXXXXX XXXXXXXXXXXXXXXXXXXXXXXXXXXX |
| | | | | | ••• |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. ^ indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.1 Food Diary. Calcium-rich Nutrients Consumption

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Visit | Time Point | Date of Assessment/ Study Day | Number of Daily Calcium Servings |
|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | XXXXXXX | Day 1 | YYYY-MM-DD/ XX | X |
| | | | Day 2 | YYYY-MM-DD/ XX | X |
| | | | Day 3 | | Not Assessed |
| | | | • • • | | |
| | | XXXXXXX | Day 1 | YYYY-MM-DD/ XX | Х |
| | | | Day 2 | YYYY-MM-DD/ XX | X |
| | | | Day 3 | YYYY-MM-DD/ XX | X |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.2 Local Skin Reactions Assessment

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Assessment | Visit | Date/ Study Day | Result | Change from Baseline |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX 14/F/A/NHL | LSR Sum Score | V1 (Day 0)<br>V2/Week2<br>V3/Week4 | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | 7 @<br>6<br>Not Done | -1 | |
| | | Investigator assessment of erosion/ulceration in lesional area | V1 (Day 0) | YYYY-MM-DD/ XX | 2 (Moderate) @ | |
| | | | V2/Week2<br>V3/Week4 | YYYY-MM-DD/ XX | 1 (Mild)<br>Not Done | |
| | | Investigator assessment of vesicles in lesional area | V1 (Day 0) | YYYY-MM-DD/ XX | 3 (Severe) @ | |
| | | | V2/Week2<br>V3/Week4 | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | 2 (Moderate)<br>2 (Moderate) | |
| | | | • • • | | | |
| | | ••• | • • • | • • • | • • • | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. LSR=Local Skin Reactions.

<sup>@</sup> indicates baseline assessment.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.3 Vital Signs

All Enrolled subjects
Page X of X

| Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter (Units) | Visit | Date of Assessment/ Study<br>Day | Result | Reference Range | Change from<br>Baseline |
|---|---|---|---|---|---|---|
| 14/F/A/NHL | Systolic Blood<br>Pressure (mm Hg) | V1 (Day0) | YYYY-MM-DD/ XX | XXX @ | XXX - XXX | |
| | _ | V2/Week2 | YYYY-MM-DD/ XX | XXX | XXX - XXX | XX |
| | | V3/Week4 | YYYY-MM-DD/ XX | XXX L | XXX - XXX | XX |
| | | • • • | ••• | • • • | • • • | • • • |
| | Diastolic Blood<br>Pressure (mm Hg) | V1 (Day0) | YYYY-MM-DD/ XX | XX @ | XXX - XXX | |
| | , 3, | V2/Week2 | YYYY-MM-DD/ XX | XX * | XXX - XXX | X |
| | | V3/Week4 | YYYY-MM-DD/ XX | XX | XXX - XXX | X |
| | | • • • | • • • | | • • • | |
| | | | • • • | | | |
| | Ethnicity | 14/F/A/NHL Systolic Blood Pressure (mm Hg) Diastolic Blood Pressure (mm Hg) | Ethnicity 14/F/A/NHL Systolic Blood Pressure (mm Hg) V2/Week2 V3/Week4 Diastolic Blood V1 (Day0) Pressure (mm Hg) V2/Week2 V3/Week4 | Ethnicity 14/F/A/NHL Systolic Blood Pressure (mm Hg) V2/Week2 YYYY-MM-DD/ XX V3/Week4 YYYY-MM-DD/ XX Diastolic Blood Pressure (mm Hg) V1 (Day0) YYYY-MM-DD/ XX V2/Week4 YYYY-MM-DD/ XX V2/Week2 YYYY-MM-DD/ XX V2/Week2 YYYY-MM-DD/ XX V3/Week4 YYYY-MM-DD/ XX V3/Week4 YYYY-MM-DD/ XX V3/Week4 YYYY-MM-DD/ XX V3/Week4 YYYY-MM-DD/ XX | ### Table | Table Tabl |

. . .

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

L = below lower reference limit. H = above upper reference limit.

<sup>@</sup> indicates baseline assessment. \* indicates notable value.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.4 Electrocardiogram

All Enrolled subjects
Page X of X

| Country/Site ID/ Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter<br>(Units) | Visit | Date of Visit/<br>Study Day | Result | Change from<br>Baseline | Findings | Comments/ Technical<br>Quality |
|---|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | General<br>Assessment | V1 (Day0) | YYYY-MM-DD/ XX | Normal @ | | | |
| | | | V3/Week4 | YYYY-MM-DD/ XX | Abnormal NCS | | XXXXXXXX; XXXXX | XXXXXXXXXXXXXX |
| | | | V5/Week8 | YYYY-MM-DD/ XX | Abnormal NCS | | | *************************************** |
| | | | • • • | • • • | • • • | • • • | | |
| | | RR Interval (msec) | V1 (Day0) | YYYY-MM-DD/ XX | XX @ | | | |
| | | | V3/Week4 | YYYY-MM-DD/ XX | XX * | XX | | |
| | | | V5/Week8 | YYYY-MM-DD/ XX | XX | XX | | |
| | | | | • • • | • • • | • • • | | |

• • •

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

L = below lower reference limit. H = above upper reference limit. CS = Clinically Significant. NCS = Not Clinically Significant.

<sup>@</sup> indicates baseline assessment. \* indicates notable value.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.5 Physical Parameters

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter (Units) | Visit | Date of Visit/ Study Day | Result | Change from Baseline |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | Weight (kg) | V1 (Day0)<br>V2/Week2<br>V3/Week4 | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | XX.X @<br>XX.X<br>XX.X | X<br>X |
| | | | | ••• | | • • • |
| | | Height (cm) | V1 (Day0)<br>V2/Week2<br>V3/Week4 | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | XXX.X @<br>XXX.X<br>XXX.X | X<br>X |
| | | | • • • | ••• | • • • | ••• |
| | | BMI (kg/m2) | | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. ^ indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.6 Physical Examination

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Examination | Visit | Date of Visit/ Study Day | Result |
|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | Abbreviated Physical Examination | Scr V1 | YYYY-MM-DD/ XX | Normal |
| | | | V1 (Day 0) | YYYY-MM-DD/ XX | Abnormal NCS |
| | | | V3/Week4 | YYYY-MM-DD/ XX | Normal |
| | | | V5/Week8 | YYYY-MM-DD/ XX | Not Done |
| | | | • • • | ••• | • • • |
| | | Complete Dermatological Examination | Scr V1 | YYYY-MM-DD/ XX | Abnormal CS |
| | | | V1 (Day 0) | YYYY-MM-DD/ XX | Normal |
| | | | V3/Week4 | YYYY-MM-DD/ XX | Normal |
| | | | V5/Week8 | YYYY-MM-DD/ XX | Normal |
| | | | • • • | ••• | • • • |
| | | | | ••• | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. CS = Clinically Significant. NCS = Not Clinically Significant.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.7 Physician Global Assessment of Psoriasis Severity

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Visit | Date/ Study Day | Result | Change from Baseline | Treatment Success |
|---|---|---|---|---|---|---|
| xxx/xx/xxxxx | 14/F/A/NHL | Scr V1<br>Scr V2<br>V1 (Day 0)<br>V2/Week2<br>V3/Week4 | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | 3 - Moderate<br>3 - Moderate<br>3 - Moderate @<br>2 - Mild<br>Not Done | -1 | |
| XXX/XX/XXXXX | 15/M/W/HL | Scr V1<br>Scr V2<br>V1 (Day 0)<br>V3/Week4<br>V5/Week | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | 3 - Moderate<br>3 - Moderate @<br>Not Done<br>0 - Clear<br>0 - Clear | -3<br>-3 | Yes<br>Yes |
| ••• | | | | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

Treatment success is defined as at least 2-point decrease from Baseline in the PGA on the trunk, limbs, and scalp.

L = below lower reference limit. H = above upper reference limit.

<sup>@</sup> indicates baseline assessment.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.8 Body Surface Area Involvement

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Parameter (Units) | Visit | Date/ Study Day | Result | Change from Baseline |
|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | Scalp BSA psoriatic involvement (%) | Scr V1<br>Scr V2<br>V1 (Day 0)<br>V3/Week4<br>V5/Week8 | YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX<br>YYYY-MM-DD/ XX | XX.X<br>XX.X<br>XX.X @<br>XX.X<br>Not Done | xx.x |
| | | Neck, Trunk and/or Limbs BSA psoriatic involvement (%) | Scr V1 Scr V2 V1 (Day 0) V3/Week4 V5/Week8 | YYYY-MM-DD/ XX YYYY-MM-DD/ XX YYYY-MM-DD/ XX YYYY-MM-DD/ XX | XX.X XX.X @ Not Done XX.X XX.X | XX.X<br>XX.X |
| | | ••• | | | | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

BSA=Body Surface Area.

<sup>@</sup> indicates baseline assessment.

 $<sup>^{\</sup>wedge}$  indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.9 Psoriasis Treatment Convenience Scale

All Enrolled subjects
Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Visit | Date/ Study Day | Parameter/Question | Score/Answe |
|---|---|---|---|---|---|
| XXX/XX/XXXX | 14/F/A/NHL | V2/Week 2 | YYYY-MM-DD/ XX | PTCS Total Score | XX |
| | | | | 1. How easy was the treatment to apply to the skin? | X |
| | | | | 2. How greasy was the treatment when applying it to the skin? | X |
| | | | | 3. How moisturized did your skin feel after applying the<br>treatment? | Not Done |
| | | • • • | | ••• | • • • |
| | | V3/Week4 | YYYY-MM-DD/ XX | PTCS Total Score | XX |
| | | | | 1. How easy was the treatment to apply to the skin? | X |
| | | | | 2. How greasy was the treatment when applying it to the skin? | X |
| | | | | 3. How moisturized did your skin feel after applying the<br>treatment? | Not Done |
| | | | | ••• | • • • |
| | | V5/Week8 | YYYY-MM-DD/ XX | PTCS Total Score | XX |
| | | | | 1. How easy was the treatment to apply to the skin? | X |
| | | | | 2. How greasy was the treatment when applying it to the skin? | X |
| | | | | 3. How moisturized did your skin feel after applying the<br>treatment? | Not Done |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male;

Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino.

PTCS=Psoriasis Treatment Convenience Scale. Question 1: From 1 = Very difficult to 10 = Very easy. Question 2: From 1 = Very greasy to 10 = Not greasy. Question 3: From 1 = Not moisturized to 10 = Very moisturized. Question 4: From 1 = Very greasy to 10 = Not greasy. Question 5: From 1 = Very disturbing to 10 = Not disturbing. Question 6: From 1 = Not satisfied to 10 = Very satisfied.

PTCS total score is the sum of the scores on questions 1 to 5.

<sup>^</sup> indicates reported visit is different from the analysis visit after windowing was performed.



MC2 Therapeutics MC2-01-C6

#### Listing 16.2.9.10 Pharmacokinetic Concentrations

All Enrolled subjects
Page X of X

| Country/Site<br>ID/ Subject<br>ID | Age (Years) / Sex/Race/ Ethnicity | Analyte | Visit | Time Point | Date, Time of Sample/<br>Study Day/ Relative Time<br>(hours) | Date, Time of Last<br>Administration of<br>Study Drug/<br>Study Day | Result | Reason if Not<br>Done |
|---|---|---|---|---|---|---|---|---|
| XXX/XX/XXXXX | 14/F/A/NHL | Betamethasone<br>17P plasma<br>concentration<br>(pg/mL) | Scr V2 | | | | XX.X | |
| | | | V2/Week2 | Pre-Dose | YYYY-MM-DD HH:MM/ XX | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | V3/Week4 | Pre-Dose | YYYY-MM-DD HH:MM/ XX (-X.XX) | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | | 1h Post-Dose | YYYY-MM-DD HH:MM/ XX (X.XX) | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | | 3h Post-Dose | YYYY-MM-DD HH:MM/ XX (X.XX) | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | | 5h Post-Dose | YYYY-MM-DD HH:MM/ XX (X.XX) | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | V5/Week8 | | YYYY-MM-DD HH:MM/ XX | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | BDP plasma<br>concentration<br>(pg/mL) | Scr V2 | | | | XX.X | |
| | | 11 31 / | V2/Week2 | Pre-Dose | YYYY-MM-DD HH:MM/ XX | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | V3/Week4 | Pre-Dose | YYYY-MM-DD HH:MM/ XX (-X.XX) | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | | 1h Post-Dose | YYYY-MM-DD HH:MM/ XX (X.XX) | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | | 3h Post-Dose | YYYY-MM-DD HH:MM/ XX (X.XX) | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | | 5h Post-Dose | YYYY-MM-DD HH:MM/ XX (X.XX) | YYYY-MM-DD HH:MM/ XX | XX.X | |
| | | | V5/Week8 | | YYYY-MM-DD HH:MM/ XX | YYYY-MM-DD HH:MM/ XX | XX.X | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. BDP=Betamethasone dipropionate; BLQ=Below Limit of Quantification.



MC2 Therapeutics MC2-01-C6

### Listing 16.2.9.11 Pharmacokinetic Parameters

PK population Page X of X

| Country/Site ID/<br>Subject ID | Age(Years)/<br>Sex/Race/<br>Ethnicity | Analyte | Parameter (Units) | Result | Reason Not Estimated |
|---|---|---|---|---|---|
| XXX/XX/XXXX | 14/F/A/NHL | BDP | Cmax (pg/mL) Tmax (h) AUCO-5 (h*pg/mL) AUCO-t (h*pg/mL) | XX.X<br>X.XX<br>NE<br>NE | XXXXXXXXXXX XXXXXXX<br>XXXXXXXXXXX XXXXXXX |
| | | Betamethasone 17-propionate | Cmax (pg/mL) Tmax (h) AUCO-5 (h*pg/mL) AUCO-t (h*pg/mL) | XX.X<br>X.XX<br>XX.X<br>XX.X | |
| | | | | ••• | |

Country: CZE=Czech Republic, HUN=Hungary, DEU=Germany; Sex: F=Female, M=Male; Race: A=Asian, B=Black or African American, W=White, O=Other; Ethnicity: HL=Hispanic or Latino, NHL=Not Hispanic or Latino. BDP=Betamethasone dipropionate, NE=Not Estimated.